CLINICAL TRIAL: NCT02453256
Title: A Phase III, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Assess the Efficacy and Safety of Tocilizumab Versus Placebo in Patients With Systemic Sclerosis
Brief Title: A Study of the Efficacy and Safety of Tocilizumab in Participants With Systemic Sclerosis (SSc)
Acronym: focuSSced
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WA29767; 2015-000424-28 (EudraCT Number)
Record Dates: First submitted 2015-05-21; First posted 2015-05-25 (Estimated); Results first posted 2019-04-03 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic | interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Double-Blind Placebo (Placebo Comparator): Participants will receive double-blind matching placebo from Baseline to Week 47. Participants may then receive open-label tocilizumab from Weeks 48 to 96.
  Interventions: Drug: Placebo; Drug: Tocilizumab
- Double-Blind Tocilizumab (Experimental): Participants will receive double-blind tocilizumab from Baseline to Week 47. Participants may then receive open-label tocilizumab from Weeks 48 to 96.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Placebo — Participants will receive matching placebo subcutaneous (SC) injections once weekly for 48 weeks of double-blind treatment.
  Arms: Double-Blind Placebo
Drug: Tocilizumab — Participants will receive 162 mg SC tocilizumab once weekly for 48 weeks of double-blind treatment. The same regimen will be given to all eligible participants for 48 weeks of open-label treatment.

SUMMARY:
This study will assess the efficacy and safety of tocilizumab compared with placebo in participants with SSc across approximately 120 planned global study sites. The study will consist of a 48-week, double-blind, placebo-controlled period followed by a 48-week open-label treatment period. Participants will be assigned, in a 1:1 ratio, to double-blind treatment with active tocilizumab or matching placebo. In the open-label period, eligible participants from either arm may receive active tocilizumab.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SSc according to American College of Rheumatology (ACR) and European League Against Rheumatism (EULAR) criteria, meeting criteria for active disease and with total disease duration of less than or equal to (</=) 60 months
* mRSS of 10-35 units, inclusive
* Agreement to remain abstinent or use an effective contraceptive method among males and females with childbearing potential

Exclusion Criteria:

* Pregnant or lactating females
* Major surgery within 8 weeks prior to screening
* Scleroderma limited to the face or areas distal to the elbows or knees
* Rheumatic autoimmune disease other than SSc
* Immunization with a live or attenuated vaccine within 4 weeks prior to Baseline
* Known hypersensitivity to human, humanized, or murine monoclonal antibodies
* Moderately severe nervous system, renal, endocrine, pulmonary, cardiovascular, or gastrointestinal (GI) disease not related to SSc, including diverticulitis or ulcerative lower GI disorders, or myocardial infarction (MI) within 6 months prior to screening
* Active or significant history of infection, including treatment with intravenous (IV) antibiotics within 4 weeks or oral antibiotics within 2 weeks prior to screening
* Significant history of tuberculosis (TB)
* Primary or secondary immunodeficiency
* Malignant disease, with the exception of excised/cured local basal or squamous cell carcinoma of the skin or carcinoma in situ of the uterine cervix
* History of drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2015-11-20 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2019-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (83):
- United States (16):
  - TriWest Research Associates, LLC, El Cajon, California
  - St. Joseph's Heritage Healthcare, Fullerton, California
  - Univ of Calif., Los Angeles; Rheumatology, Los Angeles, California
  - Arthritis Associates of Southern California, Los Angeles, California
  - Georgetown Uni. Hosp.; Rheumatology, Immunology and Allergy Dept., Washington D.C., District of Columbia
  - Rheumatology Assoc. of S. Florida - Clinical Research Center, Boca Raton, Florida
  - Millenium Research, Ormond Beach, Florida
  - Boston Univ Med Center - AC, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - West Michigan Rheumatology, PLLC, Grand Rapids, Michigan
  - Joint & Muscle Research Institute, Charlotte, North Carolina
  - Arthritis and Rheumatology; Center of Oklahoma PLLC, Oklahoma City, Oklahoma
  - Thomas Jefferson Uni ; Division of Rheumatology, Philadelphia, Pennsylvania
  - Clinical Research Center of Reading, Wyomissing, Pennsylvania
  - West Tennessee Research Institute, Jackson, Tennessee
  - Metroplex Clinical Research, Dallas, Texas
- Argentina (4):
  - Organizacion Medica de Investigacion, Buenos Aires
  - Hospital Britanico; Haematology, Buenos Aires
  - Sanatorio Parque S.A., Rosario, Santa FE
  - Centro de Investigaciones Reumatologicas Tucuman, San Miguel de Tucumán
- Belgium (2):
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
- Bulgaria (4):
  - MHAT Kaspela; Rheumatology, Plovdiv
  - MHAT-Plovdiv AD; Reumatology Department, Plovdiv
  - MHAT St.Ivan Rilski; Rheumtology Department, Sofia
  - MHAT Sv.Ivan Rilski; Clinic of Rheumatology, Sofia
- Canada (2):
  - St. Paul's Hospital University of British Colambia Division of Hematology, Vancouver, British Columbia
  - Mount Sinai Hospital; Rebecca Macdonald Centre For Arthritis & Autoimmune Disease, Toronto, Ontario
- Denmark (2):
  - Aarhus Universitetshospital Skejby, Hud- og Kønssygdomme, Aarhus N
  - Bispebjerg Hospital, Dermatologisk afdeling, København NV
- Hopital Claude Huriez; Internal Medicine, Lille, France
- Germany (5):
  - Asklepios Kllinikum Bad Abbach; Klinik für Rheumatologie und Klinische Immunologie, Bad Abbach
  - Kerckhoff-Klinik; Rheumatologie&klin.Immunologie, Bad Nauheim
  - Universitätsklinikum Dresden; Technische Universität Dresden; Rheumatologie, Innere Medizin III, Dresden
  - Klinikum der Universitat Munchen; Bereich Pettenkoferstr; Rheumaeinheit der medizinischen Klinik IV, München
  - Universitätsklinikum Tübingen Medizinische UNI-Klinik und Poliklinik Abt. Innere Medizin II, Tübingen
- Greece (2):
  - Laiko General Hospital; Dept. of Pathophysiology-Uni of Athens, Athens
  - University Hospital of Patras; Rheumatology, Pátrai
- Hungary (2):
  - National Institute of Rheumatology and Physiology, Budapest
  - Pécsi Tudományegyetem Klinikai Központ: Immunológiai és Reumatológiai Klinika, Pécs
- Italy (4):
  - Policlinico Universitario-II Università di Napoli; Reumatologia, Napoli, Campania
  - Uni ' Cattolica Del Sacro Cuore; Facoltà Di Medicina E Chirurgia A.Gemelli-Clinica Reumatologica, Rome, Lazio
  - Ospedale Maggiore Policlinico; Unità Operativa Complessa di Allergologia e Immunologia Clinica, Milan, Lombardy
  - Ospedale Careggi Villa Monnatessa ; Sezione Di Reumatologia, Florence, Tuscany
- Japan (11):
  - Gunma University Hospital, Gunma
  - Sapporo Medical University Hospital, Hokkaido
  - Hokkaido University Hospital, Hokkaido
  - Kanazawa University Hospital, Ishikawa
  - St. Marianna University School of Medicine Hospital, Kanagawa
  - Hospital of the University of Occupational and Environmental Health,Japan, Kitakyushu-shi
  - Kumamoto University Hospital, Kumamoto
  - Tohoku University Hospital, Miyagi
  - Osaka University Hospital, Osaka
  - Nippon Medical School Hospital, Tokyo
  - The University of Tokyo Hospital, Tokyo
- Lithuania (2):
  - Klaipeda University Hospital; Department of Rheumatology, Klaipėda
  - Vilnius University Hospital Santariskiu Clinic Public Insti, Vilnius
- Mexico (3):
  - Instituto Nacional de Ciencias Médicas Y de La Nutricion Zubirán, Mexico City
  - Unidad De Enfermedades; Cronico Degenerativas, SC., México
  - Cliditer SA de CV, Miexico City
- Academisch Ziekenhuis Leiden; Dept of Rheumatology, Leiden, Netherlands
- Poland (6):
  - Szpital Uniwersytecki; nr 2 im. Dr J. Biziela; Klinika Reumatologii i Ukladowych Chorob, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne; Klinika Chorob Wewnetrznych, Chorob Tkanki Łacznej i Geriatrii, Gdansk
  - Gornoslaskie Centrum Medyczne, Katowice
  - Szpital Specjalistyczny im Jozefa Dietla; Centrum Reumatologii, Immunologii i Rehabilitacji, I Oddzi, Krakow
  - SPSK NR 4; Reumatologii i Ukladowych Chorob Tkanki, Lublin
  - Narodowy Instytut Geriatrii, Reumatologii i Rehabilitacji im. Prof. Eleonory Reicher, Warsaw
- Portugal (2):
  - Hospital Garcia de Orta; Servico de Reumatologia, Almada
  - Hospital Prof. Dr. Fernando Fonseca; Medicina IV, Amadora
- Puerto Rico Clinical & Translational Research Consortium, San Juan, Puerto Rico
- Romania (2):
  - Cantacuzino Hospital; Department of Internal Medicine and Rheumatology, Bucharest
  - Spitalul Judetean Cluj; Sectia de Reumatologie, Cluj-Napoca
- Spain (3):
  - Hospital de la Santa Creu i Sant Pau; Servicio de Medicina Interna/Reumatologia, Barcelona
  - Hospital Universitario Vall d'Hebron; Servicio de Medicina Interna, Barcelona
  - Hospital General Universitario Gregorio Marañon; Servicio de Reumatología, Madrid
- Switzerland (2):
  - Universitätsspital Basel; Rheumatologische Poliklinik, Basel
  - Universitätsspital Zürich; Klinik für Rheumatologie, Zurich
- United Kingdom (6):
  - Queen Elizabeth Hospital; Rheumatology Dept., Birmingham
  - Western General Hospital, Edinburgh
  - Chapel Allerton Hospital; Leeds Institution of Rheumatology Medicine, Leeds
  - Uni Hospital Aintree; Academic Rheumatology Unit, Liverpool
  - Royal Free Hospital; Department of Rheumatology, London
  - Freeman Hospital; Musculoskeletal Unit, Newcastle upon Tyne

REFERENCES:
- [Derived] Ghuman A, Khanna D, Lin CJF, Furst DE, Raghu G, Martinez FJ, Zucchetto M, Huang S, Jennings A, Nihtyanova SI, Denton CP. Prognostic and predictive markers of systemic sclerosis-associated interstitial lung disease in a clinical trial and long-term observational cohort. Rheumatology (Oxford). 2024 Feb 1;63(2):472-481. doi: 10.1093/rheumatology/kead234. PMID 37228011
- [Derived] Khanna D, Lin CJF, Furst DE, Wagner B, Zucchetto M, Raghu G, Martinez FJ, Goldin J, Siegel J, Denton CP. Long-Term Safety and Efficacy of Tocilizumab in Early Systemic Sclerosis-Interstitial Lung Disease: Open-Label Extension of a Phase 3 Randomized Controlled Trial. Am J Respir Crit Care Med. 2022 Mar 15;205(6):674-684. doi: 10.1164/rccm.202103-0714OC. PMID 34851799
- [Derived] Roofeh D, Lin CJF, Goldin J, Kim GH, Furst DE, Denton CP, Huang S, Khanna D; focuSSced Investigators. Tocilizumab Prevents Progression of Early Systemic Sclerosis-Associated Interstitial Lung Disease. Arthritis Rheumatol. 2021 Jul;73(7):1301-1310. doi: 10.1002/art.41668. Epub 2021 May 25. PMID 33538094
- [Derived] Gao X, Jia G, Guttman A, DePianto DJ, Morshead KB, Sun KH, Ramamoorthi N, Vander Heiden JA, Modrusan Z, Wolters PJ, Jahreis A, Arron JR, Khanna D, Ramalingam TR. Osteopontin Links Myeloid Activation and Disease Progression in Systemic Sclerosis. Cell Rep Med. 2020 Nov 17;1(8):100140. doi: 10.1016/j.xcrm.2020.100140. eCollection 2020 Nov 17. PMID 33294861
- [Derived] Khanna D, Lin CJF, Furst DE, Goldin J, Kim G, Kuwana M, Allanore Y, Matucci-Cerinic M, Distler O, Shima Y, van Laar JM, Spotswood H, Wagner B, Siegel J, Jahreis A, Denton CP; focuSSced investigators. Tocilizumab in systemic sclerosis: a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Respir Med. 2020 Oct;8(10):963-974. doi: 10.1016/S2213-2600(20)30318-0. Epub 2020 Aug 28. PMID 32866440

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overall 212 participants were randomized on to the study, 107 to the placebo arm and 105 to the tocilizumab arm. One participant in placebo arm withdrew consent prior to receiving any treatment and one participant in the tocilizumab arm was withdrawn due to randomization error prior to receiving any treatment.
Groups:
- Double-Blind Placebo, Then Open Label Tocilizumab: Participants received double-blind matching placebo from Baseline to Week 48. Participants then received open-label tocilizumab from Weeks 48 to 96.
- Double-Blind Tocilizumab, Then Open Label Tocilizumab: Participants received double-blind tocilizumab from Baseline to Week 48. Participants then received open-label tocilizumab from Weeks 48 to 96.
Period: Double Blind Period
Arm/Group | Double-Blind Placebo, Then Open Label Tocilizumab | Double-Blind Tocilizumab, Then Open Label Tocilizumab
Started | 106 | 104
Completed | 93 | 95
Not Completed | 13 | 9
Not completed — Death | 1 | 1
Not completed — Adverse Event | 3 | 2
Not completed — Withdrawal by Subject | 9 | 5
Not completed — Other | 0 | 1
Period: Open Label Period
Arm/Group | Double-Blind Placebo, Then Open Label Tocilizumab | Double-Blind Tocilizumab, Then Open Label Tocilizumab
Started | 89 | 92
Completed | 82 | 85
Not Completed | 7 | 7
Not completed — Adverse Event | 1 | 3
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other | 0 | 2
Not completed — Withdrawal by Subject | 5 | 1

BASELINE CHARACTERISTICS:
Population: The analysis was conducted on the safety population, i.e. all randomized patients who received at least one dose of study drug and provided data from at least one post dose safety assessment.
Groups:
- Double-Blind Placebo, Then Tocilizumab Open Label: Participants received double-blind matching placebo from Baseline to Week 48. Participants then received open-label tocilizumab from Weeks 48 to 96.
- Double-Blind Tocilizumab, Then Tocilizumab Open Label: Participants received double-blind tocilizumab from Baseline to Week 48. Participants then received open-label tocilizumab from Weeks 48 to 96.
- Total: Total of all reporting groups
Arm/Group | Double-Blind Placebo, Then Tocilizumab Open Label | Double-Blind Tocilizumab, Then Tocilizumab Open Label | Total
Number analyzed (Participants) | 106 | 104 | 210
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.3 (12.6) | 47.0 (12.2) | 48.2 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 81 | 171
  Male | 16 | 23 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 13 | 39
  Not Hispanic or Latino | 79 | 89 | 168
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 9 | 16 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 90 | 85 | 175
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Modified Rodnan Skin Score (mRSS) During Double-blind Period
Description: The efficacy of TCZ vs placebo is evaluated in terms of in mean change in mRSS. Skin thickness will be assessed by palpation and rated using an mRSS that ranges from 0 (normal) to 3 (severe skin thickening) across 17 different body sites. The total score is the sum of the individual skin scores from all of these sites and ranges from 0 to 51 units.
Time Frame: From baseline to week 48
Population: The analysis was conducted in the Intent-to-treat (ITT) population, i.e. all patients who were randomized and received any study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Groups:
- Double-Blind Placebo: Participants received double-blind matching placebo from Baseline to Week 48. Participants may then receive open-label tocilizumab from Weeks 48 to 96.
- Double-Blind Tocilizumab: Participants received double-blind tocilizumab from Baseline to Week 48. Participants may then receive open-label tocilizumab from Weeks 48 to 96.
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 104
Units on a scale | -4.41 [-5.96 to -2.86] | -6.14 [-7.71 to -4.57]
Statistical Analysis 1: Comparison: Double-Blind Placebo vs Double-Blind Tocilizumab; Difference in least square means between the TCZ group and the Placebo group at week 48. Null hypothesis: There is no difference between the TCZ group and the placebo group in mean change in mRSS from baseline to Week 48; Test type: Superiority; p = 0.0983, Repeated Measure; Difference in least square means = -1.73, 95% CI 2-sided [-3.78 to 0.32]

2. Secondary Outcome: Percentage of Participants With Greater Than or Equal to (>/=) 20%, 40%, or 60% Improvement in mRSS During Double-blind Period
Description: The proportion of participants with threshold improvements in mRSS at Week 48 relative to baseline.
Time Frame: From Baseline to Week 48
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 104
Percentage of Participants
  ≥ 20% | 50.0 [40.01 to 59.99] | 72.1 [63.02 to 81.21]
  ≥ 40% | 37.7 [28.04 to 47.44] | 42.3 [32.33 to 52.28]
  ≥ 60% | 22.6 [14.20 to 31.08] | 17.3 [9.56 to 25.06]
Statistical Analysis 1: Comparison: Double-Blind Placebo vs Double-Blind Tocilizumab; This statistical analysis applies to participants with ≥ 20% improvement in mRSS; Test type: Superiority; p = 0.0007, Cochran-Mantel-Haenszel; Weighted difference = 21.91, 95% CI 2-sided [9.2 to 34.6]
Statistical Analysis 2: Comparison: Double-Blind Placebo vs Double-Blind Tocilizumab; This statistical analysis applies to participants with ≥ 40% improvement in mRSS; Test type: Superiority; p = 0.5139, Cochran-Mantel-Haenszel; Weighted difference = 4.32, 95% CI 2-sided [-8.7 to 17.3]
Statistical Analysis 3: Comparison: Double-Blind Placebo vs Double-Blind Tocilizumab; This statistical analysis applies to participants with ≥ 60% improvement in mRSS; Test type: Superiority; p = 0.3276, Cochran-Mantel-Haenszel; Weighted difference = -5.41, 95% CI 2-sided [-16.2 to 5.4]

3. Secondary Outcome: Change From Baseline in Percent Predicted FVC (ppFVC) During Double-blind Period
Description: FVC is pulmonary function test and will be conducted as per the study Pulmonary Function Manual, which is based on the American Thoracic Society/European Respiratory Society (ATS/ERS) Consensus Statement. FVC is the maximum amount of air exhaled from the lungs after taking the deepest breath possible. Patients perform three to eight exhalations into a spirometer with the highest value recorded.
Time Frame: Baseline to week 48
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Percent Predicted FVC
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 104
Percent Predicted FVC | -3.910 [-4.820 to -1.620] | -0.600 [-2.380 to 0.880]
Statistical Analysis 1: Comparison: Double-Blind Placebo vs Double-Blind Tocilizumab; Test type: Superiority; p = 0.0015, Van Elteren — P-value from Van Elteren analysis stratified by IL-6 level (<10; >=10 pg/mL) at screening

4. Secondary Outcome: Change in Forced Vital Capacity (FVC) During Double-blind Period
Description: as for outcome 3
Time Frame: From Baseline to Week 48
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters of air
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 104
Liters of air | -0.19 [-0.25 to -0.13] | -0.02 [-0.09 to 0.04]
Statistical Analysis 1: Comparison: Double-Blind Placebo vs Double-Blind Tocilizumab; Test type: Superiority; p = 0.0001, Repeated Measure; Difference in least square means = 0.167, 95% CI 2-sided [0.083 to 0.250]

5. Secondary Outcome: Change in Health Assessment Questionnaire Disability Index (HAQ-DI) Score During Double-blind Period
Description: The Health Assessment Questionnaire Disability Index (HAQ-DI) consists of 20 questions referring to eight component sets consisting of dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. Each item is scored on a 4-point scale from 0 to 3: 0 = Without any difficulty; 1 = With some difficulty; 2 = With much difficulty; 3 = Unable to do. Overall score was computed as the sum of component set scores and divided by the number of component sets answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty. The total score indicates the patient's self-assessed level of disability. This outcome measure represents the change in mean score from baseline. A negative change from baseline indicates improvement.
Time Frame: From Baseline to Week 48
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 104
Scores on a Scale | -0.06 [-0.16 to 0.05] | -0.11 [-0.22 to -0.01]
Statistical Analysis 1: Comparison: Double-Blind Placebo vs Double-Blind Tocilizumab; Test type: Superiority; p = 0.4489, Repeated Measure; Difference in least square means = -0.053, 95% CI 2-sided [-0.192 to 0.085]

6. Secondary Outcome: Change in Patient Global Assessment Score During Double-blind Period
Description: The Patient's Global Assessment represents the patient's overall assessment of current SSc status on a 100-mm horizontal visual analogue scale (VAS), ranging from 0 on the extreme left end of the scale indicating "has no effect at all" (symptom free), and 100 on the extreme right end indicating "worst possible effect."
Time Frame: From Baseline to Week 48
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 104
mm | -7.66 [-12.31 to -3.02] | -10.10 [-14.79 to -5.41]
Statistical Analysis 1: Comparison: Double-Blind Placebo vs Double-Blind Tocilizumab; Test type: Superiority; p = 0.4339, Repeated Measure; Difference in least square means = -2.44, 95% CI 2-sided [-8.57 to 3.70]

7. Secondary Outcome: Change in Physician Global Assessment Score During Double-blind Period
Description: The Physician's Global Assessment is to be completed on the basis of examination and overall assessment of the patient. The physician's assessment of the patient's SSc status will be scored on a 100-mm horizontal visual analogue scale (VAS), ranging from 0 on the extreme left end of the scale indicating "has no effect at all" (symptom free), and 100 on the extreme right end indicating "worst possible effect."
Time Frame: From Baseline to Week 48
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 104
mm | -19.99 [-24.76 to -15.22] | -22.45 [-27.33 to -17.57]
Statistical Analysis 1: Comparison: Double-Blind Placebo vs Double-Blind Tocilizumab; Test type: Superiority; p = 0.4378, Repeated Measure; Difference in least square means = -2.46, 95% CI 2-sided [-8.72 to 3.79]

8. Secondary Outcome: Time to Treatment Failure According to mRSS, FVC, or Protocol-Specified Event During Double-blind Period
Description: Time to treatment failure is defined as the time from randomization to the time of death, decline in percent-predicted FVC > 10% relative to baseline, > 20% increase in mRSS and an increase in mRSS of equal to or more than 5 points, or occurrence of a predefined SSc-related complication as adjudicated by the Clinical Adjudication Committee (whichever occurs first) during the 48-week double-blind treatment period. The median TTF was not estimable and is not presented for either treatment arm because of the low number of patients with events at Week 48.
Time Frame: From Baseline to Week 48
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 104
months | NA [48.7 to NA] — The median and upper limit of CI were not evaluable because of the low number of participants with events at Week 48. | NA [NA to NA] — The median, lower limit and upper limit of CI were not evaluable because of the low number of participants with events at Week 48.
Statistical Analysis 1: Comparison: Double-Blind Placebo vs Double-Blind Tocilizumab; Test type: Superiority; p = 0.0821, Cox-proportional hazards model; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.37 to 1.06]

9. Secondary Outcome: Summary of Adverse Events During Double-blind Period
Description: Summary of key safety results including Adverse Events of Special Interest (AESI). All adverse events categorized according to MedDRA version 20.1. NMSC = Non-Melanoma Skin Cancer
Time Frame: From Baseline until Week 48
Population: The analysis was conducted in the safety population i.e. received at least one dose of study drug and provide data from at least one post dose safety assessment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 104
Percentage of Participants
  At least one Adverse Event (AE) | 77.4 | 85.6
  Withdrawn from study due to an AE | 3.8 | 2.9
  Fatal AE | 2.8 | 1.0
  Serious Adverse Events (SAEs) | 17.0 | 12.5
  SAE leading to withdrawal from treatment | 3.8 | 3.8
  SAE leading to dose modification/interruption | 6.6 | 2.9
  SAE related to study drug | 6.6 | 1.0
  AE leading to withdrawal from treatment | 10.4 | 5.8
  AE leading to dose modification/interruption | 25.5 | 19.2
  AE related to study drug | 34.9 | 46.2
  Related AE leading to withdrawal from treatment | 1.9 | 1.0
  Related AE with dose modification/interruption | 16.0 | 11.5
  Infections and Infestations SAE | 6.6 | 1.9
  Infections and Infestations AE | 50.0 | 51.9
  Opportunistic Infections and Infestations AE | 0.9 | 0.0
  Malignancy AE | 0.9 | 1.9
  Malignancy AE (excluding NMSC) | 0.9 | 1.9
  At least one Hepatic SAE | 0.0 | 0.0
  At least one Stroke SAE | 0.0 | 0.0
  At least one Myocardial Infarction SAE | 1.9 | 0.0
  At least one Anaphylactic Reaction AE | 0.0 | 0.0
  Anaphylactic Reaction AE (Sampson's Criteria) | 0.0 | 0.0
  At least one Gastrointestinal Perforation SAE | 0.0 | 0.0
  At least one Bleeding SAE | 0.9 | 0.0
  At least one Demyelinating SAE | 0.0 | 0.0

10. Secondary Outcome: Incidence and Severity of Adverse Events During Double-blind Period
Description: Adverse events listed according to MedDRA version 20.1 preferred terms and severity grade.
Time Frame: From Baseline until Week 48
Population: as for outcome 9
Measure: Number; unit: Number of participants
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 104
Number of participants
  NASOPHARYNGITIS GRADE 1 | 6 | 10
  NASOPHARYNGITIS GRADE 2 | 2 | 3
  URINARY TRACT INFECTION GRADE 1 | 5 | 1
  URINARY TRACT INFECTION GRADE 2 | 5 | 3
  URINARY TRACT INFECTION GRADE 3 | 0 | 1
  GASTROENTERITIS GRADE 1 | 0 | 2
  GASTROENTERITIS GRADE 2 | 2 | 4
  HERPES ZOSTER GRADE 2 | 5 | 0
  HERPES ZOSTER GRADE 3 | 0 | 2
  PHARYNGITIS GRADE 1 | 2 | 1
  PHARYNGITIS GRADE 2 | 2 | 2
  INFECTED SKIN ULCER GRADE 1 | 0 | 1
  INFECTED SKIN ULCER GRADE 2 | 1 | 3
  INFECTED SKIN ULCER GRADE 3 | 1 | 0
  BRONCHITIS GRADE 1 | 1 | 1
  BRONCHITIS GRADE 2 | 1 | 2
  INFLUENZA GRADE 1 | 1 | 2
  INFLUENZA GRADE 2 | 1 | 1
  LATENT TUBERCULOSIS GRADE 1 | 1 | 2
  LATENT TUBERCULOSIS GRADE 2 | 0 | 2
  PNEUMONIA GRADE 2 | 1 | 1
  PNEUMONIA GRADE 3 | 3 | 0
  RESPIRATORY TRACT INFECTION GRADE 1 | 1 | 1
  RESPIRATORY TRACT INFECTION GRADE 2 | 0 | 1
  RESPIRATORY TRACT INFECTION GRADE 3 | 1 | 0
  SINUSITIS GRADE 1 | 1 | 0
  SINUSITIS GRADE 2 | 1 | 1
  SINUSITIS GRADE 3 | 0 | 1
  WOUND INFECTION GRADE 1 | 0 | 2
  WOUND INFECTION GRADE 2 | 1 | 0
  WOUND INFECTION GRADE 3 | 1 | 0
  CYSTITIS GRADE 1 | 0 | 1
  CYSTITIS GRADE 2 | 0 | 2
  LOCALISED INFECTION GRADE 1 | 1 | 0
  LOCALISED INFECTION GRADE 2 | 2 | 0
  ORAL CANDIDIASIS GRADE 1 | 2 | 1
  PARONYCHIA GRADE 2 | 2 | 0
  PARONYCHIA GRADE 3 | 1 | 0
  VULVOVAGINAL MYCOTIC INFECTION GRADE 2 | 2 | 1
  CANDIDA INFECTION GRADE 1 | 1 | 0
  CANDIDA INFECTION GRADE 2 | 1 | 0
  FOLLICULITIS GRADE 1 | 0 | 1
  FOLLICULITIS GRADE 2 | 1 | 0
  GASTROINTESTINAL INFECTION GRADE 2 | 2 | 0
  HORDEOLUM GRADE 1 | 0 | 2
  RHINITIS GRADE 2 | 1 | 1
  SOFT TISSUE INFECTION GRADE 2 | 1 | 0
  SOFT TISSUE INFECTION GRADE 4 | 1 | 0
  TINEA PEDIS GRADE 1 | 0 | 1
  TINEA PEDIS GRADE 2 | 0 | 1
  VIRAL UPPER RESPIRATORY TRACT INFECTION GRADE 1 | 1 | 0
  VIRAL UPPER RESPIRATORY TRACT INFECTION GRADE 2 | 1 | 0
  ABSCESS JAW GRADE 3 | 1 | 0
  ACUTE SINUSITIS GRADE 2 | 1 | 0
  BACTERAEMIA GRADE 2 | 1 | 0
  BODY TINEA GRADE 1 | 1 | 0
  CAMPYLOBACTER GASTROENTERITIS GRADE 1 | 0 | 1
  GASTROENTERITIS VIRAL GRADE 2 | 1 | 0
  GASTROINTESTINAL BACTERIAL OVERGROWTH GRADE 2 | 1 | 0
  GASTROINTESTINAL VIRAL INFECTION GRADE 1 | 1 | 0
  GINGIVITIS GRADE 2 | 1 | 0
  HERPES SIMPLEX GRADE 1 | 1 | 0
  INFECTIOUS MONONUCLEOSIS GRADE 1 | 1 | 0
  LARYNGITIS GRADE 1 | 1 | 0
  LICE INFESTATION GRADE 3 | 0 | 1
  OESOPHAGEAL CANDIDIASIS GRADE 2 | 1 | 0
  ORAL HERPES GRADE 2 | 1 | 0
  OSTEOMYELITIS GRADE 3 | 0 | 1
  PELVIC INFLAMMATORY DISEASE GRADE 3 | 0 | 1
  PERIODONTITIS GRADE 2 | 1 | 0
  PERIORBITAL CELLULITIS GRADE 1 | 0 | 1
  PHARYNGITIS STREPTOCOCCAL GRADE 1 | 1 | 0
  PULMONARY TUBERCULOSIS GRADE 3 | 0 | 1
  PULPITIS DENTAL GRADE 1 | 0 | 1
  PYELONEPHRITIS CHRONIC GRADE 3 | 1 | 0
  RASH PUSTULAR GRADE 1 | 0 | 1
  RESPIRATORY TRACT INFECTION BACTERIAL GRADE 2 | 0 | 1
  SEPSIS GRADE 3 | 1 | 0
  SKIN BACTERIAL INFECTION GRADE 2 | 1 | 0
  TONSILLITIS GRADE 2 | 0 | 1
  TOOTH INFECTION GRADE 3 | 1 | 0
  VIRAL INFECTION GRADE 1 | 0 | 1
  WOUND INFECTION STAPHYLOCOCCAL GRADE 1 | 0 | 1
  ARTHRALGIA GRADE 1 | 3 | 8
  ARTHRALGIA GRADE 2 | 8 | 3
  ARTHRALGIA GRADE 3 | 1 | 0
  BACK PAIN GRADE 1 | 1 | 1
  BACK PAIN GRADE 2 | 4 | 1
  MUSCLE SPASMS GRADE 1 | 1 | 2
  MUSCLE SPASMS GRADE 2 | 1 | 1
  MUSCLE SPASMS GRADE 3 | 1 | 0
  PAIN IN EXTREMITY GRADE 1 | 2 | 2
  PAIN IN EXTREMITY GRADE 2 | 0 | 1
  PAIN IN EXTREMITY GRADE 3 | 1 | 0
  MUSCULOSKELETAL PAIN GRADE 1 | 1 | 0
  MUSCULOSKELETAL PAIN GRADE 2 | 4 | 0
  BURSITIS GRADE 1 | 3 | 0
  BURSITIS GRADE 2 | 0 | 1
  MYALGIA GRADE 1 | 1 | 0
  MYALGIA GRADE 2 | 3 | 0
  ARTHRITIS GRADE 2 | 2 | 1
  INTERVERTEBRAL DISC PROTRUSION GRADE 1 | 1 | 1
  INTERVERTEBRAL DISC PROTRUSION GRADE 2 | 0 | 1
  MYOSITIS GRADE 1 | 1 | 0
  MYOSITIS GRADE 2 | 1 | 1
  OSTEOCHONDROSIS GRADE 1 | 1 | 2
  FOOT DEFORMITY GRADE 1 | 1 | 1
  SCLERODERMA GRADE 2 | 0 | 1
  SCLERODERMA GRADE 4 | 1 | 0
  SJOGREN'S SYNDROME GRADE 1 | 1 | 0
  SJOGREN'S SYNDROME GRADE 2 | 1 | 0
  SPINAL OSTEOARTHRITIS GRADE 1 | 0 | 1
  SPINAL OSTEOARTHRITIS GRADE 2 | 1 | 0
  EXTREMITY CONTRACTURE GRADE 1 | 1 | 0
  FIBROMYALGIA GRADE 1 | 1 | 0
  FLANK PAIN GRADE 1 | 0 | 1
  JOINT STIFFNESS GRADE 1 | 0 | 1
  JOINT SWELLING GRADE 2 | 1 | 0
  MUSCLE CONTRACTURE GRADE 1 | 0 | 1
  MUSCLE FATIGUE GRADE 1 | 1 | 0
  MUSCULAR WEAKNESS GRADE 2 | 0 | 1
  MUSCULOSKELETAL CHEST PAIN GRADE 1 | 1 | 0
  MYOPATHY GRADE 1 | 1 | 0
  NECK PAIN GRADE 2 | 1 | 0
  OSTEOPENIA GRADE 1 | 0 | 1
  OSTEOPOROSIS GRADE 2 | 0 | 1
  OSTEOPOROTIC FRACTURE GRADE 2 | 1 | 0
  PAIN IN JAW GRADE 1 | 1 | 0
  POLYARTHRITIS GRADE 2 | 1 | 0
  TENOSYNOVITIS GRADE 2 | 0 | 1
  TENOSYNOVITIS STENOSANS GRADE 1 | 1 | 0
  SKIN ULCER GRADE 1 | 5 | 8
  SKIN ULCER GRADE 2 | 7 | 5
  SKIN ULCER GRADE 3 | 0 | 2
  PRURITUS GRADE 1 | 2 | 1
  PRURITUS GRADE 2 | 2 | 5
  RASH GRADE 1 | 4 | 2
  RASH GRADE 2 | 3 | 0
  ERYTHEMA GRADE 1 | 1 | 4
  ECZEMA GRADE 1 | 0 | 2
  ECZEMA GRADE 2 | 2 | 0
  ROSACEA GRADE 1 | 0 | 1
  ROSACEA GRADE 2 | 1 | 1
  SKIN TIGHTNESS GRADE 1 | 2 | 1
  DERMATITIS CONTACT GRADE 2 | 1 | 1
  INGROWING NAIL GRADE 1 | 0 | 1
  INGROWING NAIL GRADE 2 | 1 | 0
  MACULE GRADE 1 | 1 | 1
  NIGHT SWEATS GRADE 1 | 2 | 0
  SKIN DISCOLOURATION GRADE 1 | 0 | 2
  SKIN FISSURES GRADE 1 | 0 | 2
  SKIN HYPERTROPHY GRADE 1 | 0 | 2
  SKIN INDURATION GRADE 1 | 2 | 0
  URTICARIA GRADE 1 | 0 | 1
  URTICARIA GRADE 2 | 1 | 0
  ALOPECIA GRADE 1 | 0 | 1
  BLISTER GRADE 2 | 0 | 1
  CHLOASMA GRADE 1 | 1 | 0
  COLD SWEAT GRADE 1 | 1 | 0
  DECUBITUS ULCER GRADE 2 | 0 | 1
  DERMATITIS ACNEIFORM GRADE 1 | 0 | 1
  DERMATITIS ATOPIC GRADE 1 | 0 | 1
  DIGITAL PITTING SCAR GRADE 4 | 1 | 0
  DRY SKIN GRADE 1 | 0 | 1
  ECCHYMOSIS GRADE 3 | 1 | 0
  EXCESSIVE GRANULATION TISSUE GRADE 3 | 0 | 1
  HYPERTRICHOSIS GRADE 1 | 1 | 0
  ONYCHOLYSIS GRADE 1 | 1 | 0
  PAIN OF SKIN GRADE 1 | 1 | 0
  PAPULE GRADE 1 | 1 | 0
  RASH ERYTHEMATOUS GRADE 1 | 0 | 1
  RASH MACULO-PAPULAR GRADE 3 | 0 | 1
  SKIN DEPIGMENTATION GRADE 1 | 1 | 0
  SKIN FIBROSIS GRADE 2 | 1 | 0
  SKIN HYPOPIGMENTATION GRADE 1 | 1 | 0
  SKIN OEDEMA GRADE 1 | 1 | 0
  VITILIGO GRADE 2 | 1 | 0
  DIARRHOEA GRADE 1 | 5 | 6
  DIARRHOEA GRADE 2 | 3 | 0
  GASTROOESOPHAGEAL REFLUX DISEASE GRADE 1 | 3 | 3
  GASTROOESOPHAGEAL REFLUX DISEASE GRADE 2 | 2 | 1
  NAUSEA GRADE 1 | 5 | 3
  NAUSEA GRADE 2 | 1 | 0
  ABDOMINAL PAIN GRADE 1 | 3 | 1
  ABDOMINAL PAIN GRADE 2 | 1 | 0
  ABDOMINAL PAIN GRADE 3 | 1 | 0
  CONSTIPATION GRADE 1 | 2 | 2
  CONSTIPATION GRADE 2 | 2 | 0
  DYSPEPSIA GRADE 1 | 1 | 2
  DYSPEPSIA GRADE 2 | 1 | 1
  DYSPHAGIA GRADE 1 | 2 | 2
  DYSPHAGIA GRADE 2 | 0 | 1
  STOMATITIS GRADE 1 | 1 | 1
  STOMATITIS GRADE 2 | 1 | 0
  VOMITING GRADE 1 | 1 | 1
  VOMITING GRADE 3 | 0 | 1
  ABDOMINAL DISCOMFORT GRADE 1 | 0 | 1
  ABDOMINAL DISCOMFORT GRADE 2 | 1 | 0
  ABDOMINAL DISTENSION GRADE 1 | 1 | 0
  ABDOMINAL DISTENSION GRADE 2 | 1 | 0
  ABDOMINAL PAIN UPPER GRADE 1 | 1 | 1
  DENTAL CARIES GRADE 2 | 1 | 1
  FAECES SOFT GRADE 1 | 1 | 1
  HAEMORRHOIDS GRADE 1 | 1 | 0
  HAEMORRHOIDS GRADE 2 | 1 | 0
  TOOTHACHE GRADE 2 | 2 | 0
  ANAL HAEMORRHAGE GRADE 2 | 1 | 0
  CHRONIC GASTRITIS GRADE 1 | 1 | 0
  DIVERTICULUM INTESTINAL GRADE 1 | 0 | 1
  DRY MOUTH GRADE 2 | 0 | 1
  DUODENITIS GRADE 1 | 0 | 1
  GASTRIC DISORDER GRADE 1 | 0 | 1
  GASTRIC POLYPS GRADE 1 | 1 | 0
  GASTRITIS GRADE 2 | 1 | 0
  HAEMATOCHEZIA GRADE 1 | 0 | 1
  ILEUS PARALYTIC GRADE 3 | 1 | 0
  LOOSE TOOTH GRADE 1 | 0 | 1
  OESOPHAGEAL DISORDER GRADE 1 | 1 | 0
  OESOPHAGEAL HYPOMOTILITY GRADE 2 | 0 | 1
  PERIODONTAL DISEASE GRADE 2 | 1 | 0
  PNEUMATOSIS INTESTINALIS GRADE 2 | 0 | 1
  RANULA GRADE 1 | 0 | 1
  SWOLLEN TONGUE GRADE 2 | 0 | 1
  FATIGUE GRADE 1 | 3 | 7
  FATIGUE GRADE 2 | 4 | 1
  OEDEMA PERIPHERAL GRADE 1 | 2 | 1
  OEDEMA PERIPHERAL GRADE 2 | 1 | 0
  ASTHENIA GRADE 1 | 2 | 0
  ASTHENIA GRADE 3 | 1 | 0
  CALCINOSIS GRADE 1 | 1 | 2
  INJECTION SITE ERYTHEMA GRADE 1 | 0 | 1
  INJECTION SITE ERYTHEMA GRADE 2 | 0 | 1
  INJECTION SITE ERYTHEMA GRADE 3 | 0 | 1
  INJECTION SITE REACTION GRADE 1 | 0 | 1
  INJECTION SITE REACTION GRADE 2 | 1 | 1
  PAIN GRADE 2 | 1 | 0
  PAIN GRADE 3 | 0 | 1
  PAIN GRADE 4 | 1 | 0
  CHEST PAIN GRADE 1 | 2 | 0
  CYST GRADE 1 | 1 | 0
  CYST GRADE 2 | 1 | 0
  INFLUENZA LIKE ILLNESS GRADE 1 | 1 | 1
  DEATH GRADE 5 | 0 | 1
  FEELING HOT GRADE 1 | 0 | 1
  GRANULOMA GRADE 1 | 1 | 0
  INJECTION SITE EXTRAVASATION GRADE 1 | 0 | 1
  INJECTION SITE INDURATION GRADE 2 | 0 | 1
  INJECTION SITE PRURITUS GRADE 2 | 0 | 1
  MALAISE GRADE 1 | 0 | 1
  NODULE GRADE 1 | 1 | 0
  PERIPHERAL SWELLING GRADE 2 | 1 | 0
  PYREXIA GRADE 1 | 1 | 0
  SENSATION OF FOREIGN BODY GRADE 1 | 0 | 1
  VESSEL PUNCTURE SITE PAIN GRADE 1 | 0 | 1
  WEIGHT DECREASED GRADE 1 | 3 | 1
  WEIGHT DECREASED GRADE 2 | 3 | 2
  ALANINE AMINOTRANSFERASE INCREASED GRADE 1 | 0 | 2
  ALANINE AMINOTRANSFERASE INCREASED GRADE 2 | 2 | 0
  ALANINE AMINOTRANSFERASE INCREASED GRADE 3 | 0 | 2
  ASPARTATE AMINOTRANSFERASE INCREASED GRADE 1 | 0 | 2
  ASPARTATE AMINOTRANSFERASE INCREASED GRADE 2 | 2 | 0
  ASPARTATE AMINOTRANSFERASE INCREASED GRADE 3 | 0 | 1
  HEPATIC ENZYME INCREASED GRADE 1 | 1 | 0
  HEPATIC ENZYME INCREASED GRADE 2 | 1 | 1
  HEPATIC ENZYME INCREASED GRADE 3 | 1 | 0
  WEIGHT INCREASED GRADE 1 | 2 | 2
  TRANSAMINASES INCREASED GRADE 1 | 0 | 1
  TRANSAMINASES INCREASED GRADE 2 | 2 | 0
  BLOOD CHOLESTEROL INCREASED GRADE 1 | 0 | 1
  BLOOD CHOLESTEROL INCREASED GRADE 2 | 0 | 1
  UPPER RESPIRATORY TRACT INFECTION GRADE 1 | 4 | 7
  UPPER RESPIRATORY TRACT INFECTION GRADE 2 | 7 | 4
  UPPER RESPIRATORY TRACT INFECTION GRADE 3 | 0 | 1
  BLOOD CREATINE PHOSPHOKINASE INCREASED GRADE 1 | 0 | 1
  BLOOD CREATINE PHOSPHOKINASE INCREASED GRADE 2 | 0 | 1
  BLOOD BILIRUBIN INCREASED GRADE 1 | 0 | 1
  BLOOD URINE PRESENT GRADE 2 | 1 | 0
  CAROTID INTIMA-MEDIA THICKNESS INCREASED GRADE 1 | 1 | 0
  COMPUTERISED TOMOGRAM THORAX ABNORMAL GRADE 2 | 1 | 0
  HAEMOGLOBIN DECREASED GRADE 2 | 1 | 0
  LIVER FUNCTION TEST ABNORMAL GRADE 2 | 0 | 1
  LOW DENSITY LIPOPROTEIN INCREASED GRADE 2 | 0 | 1
  PROTEIN URINE PRESENT GRADE 2 | 1 | 0
  TRANSFERRIN SATURATION INCREASED GRADE 1 | 0 | 1
  TUBERCULIN TEST POSITIVE GRADE 2 | 1 | 0
  URINE BILIRUBIN INCREASED GRADE 2 | 1 | 0
  UROBILINOGEN URINE INCREASED GRADE 2 | 1 | 0
  WHITE BLOOD CELLS URINE POSITIVE GRADE 1 | 1 | 0
  COUGH GRADE 1 | 3 | 1
  COUGH GRADE 2 | 2 | 2
  INTERSTITIAL LUNG DISEASE GRADE 1 | 3 | 0
  INTERSTITIAL LUNG DISEASE GRADE 2 | 5 | 0
  DYSPNOEA GRADE 1 | 1 | 1
  DYSPNOEA GRADE 2 | 2 | 2
  EPISTAXIS GRADE 1 | 3 | 1
  EPISTAXIS GRADE 2 | 0 | 1
  DYSPNOEA EXERTIONAL GRADE 1 | 1 | 0
  DYSPNOEA EXERTIONAL GRADE 2 | 1 | 0
  DYSPNOEA EXERTIONAL GRADE 3 | 1 | 0
  OROPHARYNGEAL PAIN GRADE 1 | 1 | 1
  OROPHARYNGEAL PAIN GRADE 2 | 1 | 0
  PRODUCTIVE COUGH GRADE 1 | 2 | 0
  DYSPHONIA GRADE 1 | 1 | 0
  HAEMOPTYSIS GRADE 1 | 0 | 1
  PAINFUL RESPIRATION GRADE 1 | 1 | 0
  PLEURAL EFFUSION GRADE 4 | 1 | 0
  PNEUMONITIS GRADE 2 | 1 | 0
  RHINITIS ALLERGIC GRADE 1 | 1 | 0
  RHINORRHOEA GRADE 1 | 1 | 0
  HEADACHE GRADE 1 | 3 | 3
  HEADACHE GRADE 2 | 4 | 0
  DIZZINESS GRADE 1 | 2 | 2
  DIZZINESS GRADE 2 | 1 | 1
  NEUROPATHY PERIPHERAL GRADE 2 | 2 | 0
  POST HERPETIC NEURALGIA GRADE 2 | 2 | 0
  CARPAL TUNNEL SYNDROME GRADE 1 | 1 | 0
  DYSGEUSIA GRADE 1 | 1 | 0
  HYPOAESTHESIA GRADE 1 | 1 | 0
  HYPOKINESIA GRADE 3 | 0 | 1
  MEMORY IMPAIRMENT GRADE 1 | 0 | 1
  NERVE COMPRESSION GRADE 1 | 1 | 0
  NEURALGIA GRADE 1 | 1 | 0
  PARAESTHESIA GRADE 1 | 0 | 1
  PARKINSONISM GRADE 2 | 1 | 0
  PRESYNCOPE GRADE 1 | 0 | 1
  RADICULAR PAIN GRADE 1 | 0 | 1
  SENSORY LOSS GRADE 1 | 1 | 0
  SOMNOLENCE GRADE 1 | 0 | 1
  LIMB INJURY GRADE 1 | 2 | 1
  LIMB INJURY GRADE 2 | 2 | 0
  LIMB INJURY GRADE 3 | 0 | 1
  FALL GRADE 1 | 0 | 1
  FALL GRADE 2 | 0 | 2
  EAR INJURY GRADE 1 | 0 | 2
  LACERATION GRADE 1 | 1 | 0
  LACERATION GRADE 2 | 1 | 0
  SCAR GRADE 1 | 0 | 1
  SCAR GRADE 2 | 1 | 0
  WOUND GRADE 1 | 0 | 1
  WOUND GRADE 2 | 1 | 0
  ANIMAL BITE GRADE 2 | 0 | 1
  ANKLE FRACTURE GRADE 1 | 0 | 1
  ARTHROPOD STING GRADE 1 | 1 | 0
  CONTUSION GRADE 1 | 0 | 1
  CRANIOCEREBRAL INJURY GRADE 2 | 1 | 0
  EXCORIATION GRADE 1 | 0 | 1
  FACE INJURY GRADE 1 | 0 | 1
  INJURY CORNEAL GRADE 2 | 1 | 0
  JOINT INJURY GRADE 3 | 0 | 1
  LIGAMENT SPRAIN GRADE 1 | 0 | 1
  LIMB TRAUMATIC AMPUTATION GRADE 3 | 0 | 1
  MENISCUS INJURY GRADE 3 | 0 | 1
  MUSCLE RUPTURE GRADE 2 | 0 | 1
  MUSCLE STRAIN GRADE 2 | 1 | 0
  ROAD TRAFFIC ACCIDENT GRADE 1 | 0 | 1
  SKIN ABRASION GRADE 1 | 1 | 0
  SPINAL COMPRESSION FRACTURE GRADE 2 | 1 | 0
  THERMAL BURN GRADE 1 | 0 | 1
  ANAEMIA GRADE 1 | 3 | 0
  ANAEMIA GRADE 2 | 2 | 1
  ANAEMIA GRADE 3 | 1 | 0
  IRON DEFICIENCY ANAEMIA GRADE 1 | 1 | 0
  IRON DEFICIENCY ANAEMIA GRADE 2 | 1 | 0
  IRON DEFICIENCY ANAEMIA GRADE 3 | 0 | 1
  LYMPHOPENIA GRADE 2 | 0 | 1
  LYMPHOPENIA GRADE 3 | 1 | 0
  NEUTROPENIA GRADE 2 | 0 | 1
  NEUTROPENIA GRADE 3 | 1 | 0
  ANAEMIA MEGALOBLASTIC GRADE 2 | 1 | 0
  EOSINOPHILIA GRADE 1 | 0 | 1
  LEUKOCYTOSIS GRADE 1 | 1 | 0
  LEUKOPENIA GRADE 2 | 0 | 1
  LYMPHADENOPATHY MEDIASTINAL GRADE 2 | 1 | 0
  MICROANGIOPATHIC HAEMOLYTIC ANAEMIA GRADE 2 | 0 | 1
  MICROCYTIC ANAEMIA GRADE 1 | 0 | 1
  THROMBOCYTOPENIA GRADE 1 | 0 | 1
  DECREASED APPETITE GRADE 1 | 4 | 1
  DYSLIPIDAEMIA GRADE 1 | 0 | 2
  DYSLIPIDAEMIA GRADE 2 | 1 | 1
  HYPERCHOLESTEROLAEMIA GRADE 1 | 0 | 1
  HYPERCHOLESTEROLAEMIA GRADE 2 | 0 | 1
  HYPERTRIGLYCERIDAEMIA GRADE 2 | 1 | 1
  DIABETES MELLITUS GRADE 2 | 1 | 0
  DIABETIC KETOACIDOSIS GRADE 4 | 1 | 0
  DIABETIC METABOLIC DECOMPENSATION GRADE 1 | 0 | 1
  FOLATE DEFICIENCY GRADE 1 | 0 | 1
  GOUT GRADE 2 | 1 | 0
  HYPERGLYCAEMIA GRADE 3 | 1 | 0
  HYPERLIPIDAEMIA GRADE 1 | 0 | 1
  HYPONATRAEMIA GRADE 1 | 1 | 0
  IRON DEFICIENCY GRADE 2 | 1 | 0
  OBESITY GRADE 1 | 0 | 1
  WEIGHT FLUCTUATION GRADE 1 | 1 | 0
  PALPITATIONS GRADE 1 | 4 | 1
  PALPITATIONS GRADE 3 | 0 | 1
  BUNDLE BRANCH BLOCK RIGHT GRADE 1 | 1 | 0
  BUNDLE BRANCH BLOCK RIGHT GRADE 2 | 0 | 1
  PERICARDIAL EFFUSION GRADE 1 | 1 | 0
  PERICARDIAL EFFUSION GRADE 2 | 1 | 0
  ACUTE MYOCARDIAL INFARCTION GRADE 3 | 1 | 0
  ANGINA PECTORIS GRADE 3 | 0 | 1
  ATRIAL FIBRILLATION GRADE 3 | 1 | 0
  ATRIAL TACHYCARDIA GRADE 2 | 1 | 0
  BRADYCARDIA GRADE 1 | 0 | 1
  CARDIAC FAILURE GRADE 3 | 0 | 1
  CARDIAC FAILURE CHRONIC GRADE 5 | 1 | 0
  MICROVASCULAR CORONARY ARTERY DISEASE GRADE 2 | 1 | 0
  MYOCARDIAL INFARCTION GRADE 5 | 1 | 0
  MYOCARDITIS GRADE 5 | 1 | 0
  PERICARDITIS GRADE 2 | 1 | 0
  SUPRAVENTRICULAR EXTRASYSTOLES GRADE 1 | 1 | 0
  TACHYCARDIA GRADE 1 | 1 | 0
  ANXIETY GRADE 1 | 2 | 1
  ANXIETY GRADE 2 | 1 | 0
  INSOMNIA GRADE 1 | 2 | 1
  STRESS GRADE 1 | 1 | 1
  ADJUSTMENT DISORDER GRADE 3 | 1 | 0
  DEPRESSED MOOD GRADE 3 | 0 | 1
  DEPRESSION GRADE 1 | 0 | 1
  GENERALISED ANXIETY DISORDER GRADE 2 | 1 | 0
  SLEEP DISORDER GRADE 1 | 1 | 0
  CHALAZION GRADE 1 | 0 | 2
  GLAUCOMA GRADE 1 | 0 | 1
  GLAUCOMA GRADE 3 | 1 | 0
  BLEPHARITIS GRADE 2 | 0 | 1
  CATARACT GRADE 3 | 1 | 0
  CONJUNCTIVAL HAEMORRHAGE GRADE 1 | 1 | 0
  DRY EYE GRADE 1 | 0 | 1
  EYELID OEDEMA GRADE 1 | 0 | 1
  KERATITIS GRADE 2 | 0 | 1
  VISUAL IMPAIRMENT GRADE 1 | 0 | 1
  RAYNAUD'S PHENOMENON GRADE 1 | 1 | 3
  RAYNAUD'S PHENOMENON GRADE 2 | 1 | 0
  BLOOD PRESSURE FLUCTUATION GRADE 1 | 0 | 1
  HYPERTENSION GRADE 2 | 0 | 1
  HYPOTENSION GRADE 2 | 1 | 0
  PERIPHERAL ISCHAEMIA GRADE 2 | 0 | 1
  THROMBOPHLEBITIS GRADE 2 | 0 | 1
  VASCULITIS GRADE 2 | 1 | 0
  ACUTE KIDNEY INJURY GRADE 3 | 1 | 0
  DYSURIA GRADE 1 | 1 | 0
  HAEMATURIA GRADE 1 | 1 | 0
  NEPHROLITHIASIS GRADE 3 | 0 | 1
  RENAL COLIC GRADE 2 | 0 | 1
  RENAL CYST GRADE 1 | 1 | 0
  RENAL PAIN GRADE 2 | 1 | 0
  SCLERODERMA RENAL CRISIS GRADE 3 | 0 | 1
  AMENORRHOEA GRADE 1 | 0 | 1
  BREAST CYST GRADE 1 | 1 | 0
  CERVICAL POLYP GRADE 1 | 0 | 1
  ERECTILE DYSFUNCTION GRADE 2 | 1 | 0
  GENITAL RASH GRADE 2 | 1 | 0
  MENSTRUATION IRREGULAR GRADE 1 | 1 | 0
  OVARIAN CYST RUPTURED GRADE 2 | 1 | 0
  PENILE PAIN GRADE 1 | 1 | 0
  B-CELL LYMPHOMA GRADE 3 | 0 | 1
  BENIGN BONE NEOPLASM GRADE 3 | 1 | 0
  BENIGN LUNG NEOPLASM GRADE 1 | 0 | 1
  BREAST CANCER GRADE 3 | 0 | 1
  LUNG ADENOCARCINOMA GRADE 4 | 1 | 0
  SKIN PAPILLOMA GRADE 2 | 0 | 1
  FOOD ALLERGY GRADE 2 | 0 | 1
  HYPERSENSITIVITY GRADE 1 | 0 | 1
  TYPE I HYPERSENSITIVITY GRADE 2 | 0 | 1
  MICROSTOMIA GRADE 1 | 1 | 0
  MICROSTOMIA GRADE 2 | 0 | 1
  PRESBYACUSIS GRADE 1 | 0 | 1
  VERTIGO GRADE 1 | 1 | 0
  HYPOTHYROIDISM GRADE 1 | 0 | 1
  THYROID MASS GRADE 1 | 1 | 0
  HEPATIC STEATOSIS GRADE 1 | 0 | 1
  NEEDLE ISSUE GRADE 1 | 0 | 1
  CATARACT OPERATION GRADE 3 | 1 | 0

11. Secondary Outcome: Number of Participants With Adverse Events Leading to Death During Double-blind Period
Description: Reason of death is coded using MedDRA 20.1
Time Frame: From Baseline up to Week 48
Population: as for outcome 9
Measure: Number; unit: Number of participants
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 104
Number of participants
  CARDIAC FAILURE CHRONIC | 1 | 0
  MYOCARDITIS | 1 | 0
  MYOCARDIAL INFARCTION | 1 | 0
  DEATH | 0 | 1

12. Secondary Outcome: Frequency of Serious Systemic Sclerosis (SSC) Related Complications During Double-blind Period
Description: Adverse event terms coded using MedDRA 20.1. Includes only those serious events adjudicated as SSC-related complications by an independent external committee.
Time Frame: From Baseline up to Week 48
Population: as for outcome 9
Measure: Number; unit: Number of Participants
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 104
Number of Participants
  CARDIAC FAILURE | 0 | 1
  CARDIAC FAILURE CHRONIC | 1 | 0
  MICROVASCULAR CORONARY ARTERY DISEASE | 1 | 0
  MYOCARDITIS | 1 | 0
  INFECTED SKIN ULCER | 1 | 0
  OSTEOMYELITIS | 0 | 1
  WOUND INFECTION | 0 | 1
  ILEUS PARALYTIC | 1 | 0
  PAIN | 1 | 0
  WEIGHT DECREASED | 0 | 1
  SCLERODERMA | 1 | 0
  HYPOKINESIA | 0 | 1
  ADJUSTMENT DISORDER | 1 | 0
  SCLERODERMA RENAL CRISIS | 0 | 1
  DIGITAL PITTING SCAR | 1 | 0

13. Secondary Outcome: Incidence of Haematology and Hepatic Laboratory Parameters During Double-blind Period
Description: A laboratory event occurred if the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) grade for a post-baseline laboratory measurement increased from baseline.
Time Frame: From Baseline up to Week 48
Population: as for outcome 9
Measure: Number; unit: Number of Participants
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 104
Number of Participants
  High Alkaline Phosphatase | 7 | 1
  High SGPT/ALT | 17 | 32
  High SGOT/AST | 17 | 24
  Low Neutrophils, Segmented, Abs | 2 | 27
  Low Platelet | 0 | 9
  High Bilirubin | 1 | 13

14. Secondary Outcome: Percentage of Participants With Change in Digital Ulcer Count During Double-blind Period
Description: A digital ulcer is defined as an ulcer at or distal to the MCP joint on either the dorsal or volar surface, with loss of surface epithelialization. This does not include fissures, cracks, or calcium extrusions from calcinosis cutis. The number of fingers (0-10) with digital ulcers and the number of digital (or finger) ulcers will be counted and recorded by the investigator.
Time Frame: From Baseline to Week 48
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 104
Percentage of participants
  No change | 85.4 | 87.2
  Increase by 1 | 3.4 | 5.3
  Increase by 2 | 1.1 | 1.1
  Increase by 3 | 0 | 0
  Increase by 4 | 0 | 0
  Increase by >4 | 1.1 | 0
  Decrease by 1 | 3.4 | 4.3
  Decrease by 2 | 3.4 | 0
  Decrease by 3 | 0 | 1.1
  Decrease by 4 | 1.1 | 0
  Decrease by >4 | 0 | 0
  Baseline missing | 1.1 | 1.1

15. Secondary Outcome: Percentage of Participants With Positive Anti-Tocilizumab Assay Result at Baseline
Description: Incidence of anti-Tocilizumab at baseline
Time Frame: Baseline
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 104
Percentage of Participants | 5.9 | 2.9

16. Secondary Outcome: Percentage of Participants With Positive Anti-Tocilizumab Assay Post-Baseline up to Week 48
Description: Incidence of anti-Tocilizumab antibodies during the study relative to the prevalence of anti-Tocilizumab antibodies at baseline. Samples that are positive for anti-TCZ in the screening assay will be further analyzed by a confirmation assay to confirm specificity. If the confirmation assay is positive, two additional tests will be performed: a neutralizing assay for the ability to inhibit the activity of TCZ and a test for anti -TCZ of the IgE isotype.
Time Frame: Double-blind period (up to Week 48)
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 104
Percentage of Participants
  Positive Anti-TCZ Assay: number analyzed (Participants) | 101 | 104
  Positive Anti-TCZ Assay | 0.0 | 2.9
  Positive Confirmation Assay: number analyzed (Participants) | 101 | 104
  Positive Confirmation Assay | 0.0 | 1.0
  Positive Neutralizing Assay: number analyzed (Participants) | 101 | 104
  Positive Neutralizing Assay | 0.0 | 1.0
  Positive IgE Assay: number analyzed (Participants) | 101 | 104
  Positive IgE Assay | 0.0 | 0.0

17. Secondary Outcome: Correlation Between Anti-Tocilizumab Antibody Status and Outcome Measures Pertaining to the Efficacy, Safety, and Pharmacokinetics of Tocilizumab
Description: Pre-specified analysis of the relationship between Anti-Tocilizumab Antibody status and safety, efficacy, and PK endpoints were not analyzed via subgroup analyses as there was only 1 patient with ADA-positive status.
Time Frame: Baseline; during Weeks 8, 16, 24, 36, 48, 96, and/or at treatment discontinuation (up to 96 weeks); and 8 weeks after treatment discontinuation (up to 104 weeks overall)
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 104
Units on a scale | NA [NA to NA] — Pre-specified analysis of the relationship between Anti-Tocilizumab Antibody status and safety, efficacy, and PK endpoints were not analyzed via subgroup analyses as there was only 1 patient with ADA-positive status. | NA [NA to NA] — Pre-specified analysis of the relationship between Anti-Tocilizumab Antibody status and safety, efficacy, and PK endpoints were not analyzed via subgroup analyses as there was only 1 patient with ADA-positive status.

18. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR), Mean, From Baseline to Week 48
Description: Erythrocyte Sedimentation Rate (ESR) levels predose at baseline and at subsequent time points after initiation of study drug.
Time Frame: From Predose up to Week 48
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 104
mm/hr
  Baseline: number analyzed (Participants) | 103 | 100
  Baseline | 34.72 (18.49) | 34.83 (16.29)
  Week 4: number analyzed (Participants) | 96 | 98
  Week 4 | 31.38 (19.00) | 14.29 (12.98)
  Week 24: number analyzed (Participants) | 98 | 94
  Week 24 | 28.49 (20.86) | 8.46 (8.63)
  Week 48: number analyzed (Participants) | 88 | 90
  Week 48 | 26.59 (18.62) | 10.82 (15.53)

19. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR), Median, From Baseline to Week 48
Description: as for outcome 18
Time Frame: From Baseline to Week 48
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: mm/hr
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 104
mm/hr
  Baseline: number analyzed (Participants) | 103 | 100
  Baseline | 33.0 [23.00 to 43.00] | 33.50 [26.00 to 42.00]
  Week 4: number analyzed (Participants) | 96 | 98
  Week 4 | 30.00 [16.50 to 39.50] | 9.50 [4.00 to 23.00]
  Week 24: number analyzed (Participants) | 98 | 94
  Week 24 | 25.00 [12.00 to 36.00] | 5.00 [3.00 to 8.00]
  Week 48: number analyzed (Participants) | 88 | 90
  Week 48 | 22.50 [14.00 to 31.50] | 5.50 [3.00 to 12.00]

20. Secondary Outcome: Serum Interleukin (IL)-6 Level, Mean, From Baseline to Week 48
Description: Serum Interleukin (IL)-6 levels predose at baseline and at subsequent time points after initiation of study drug.
Time Frame: From Baseline to Week 48
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 104
pg/mL
  Baseline | 11.83 (19.74) | 13.88 (43.77)
  Week 4: number analyzed (Participants) | 95 | 99
  Week 4 | 13.41 (29.98) | 143.97 (427.01)
  Week 8: number analyzed (Participants) | 95 | 94
  Week 8 | 14.21 (26.82) | 111.44 (280.34)
  Week 16: number analyzed (Participants) | 93 | 88
  Week 16 | 15.40 (24.26) | 66.20 (70.50)
  Week 24: number analyzed (Participants) | 85 | 85
  Week 24 | 11.81 (24.05) | 62.74 (53.40)
  Week 36: number analyzed (Participants) | 73 | 83
  Week 36 | 9.32 (15.23) | 62.15 (68.08)
  Week 48: number analyzed (Participants) | 78 | 80
  Week 48 | 9.25 (15.14) | 53.98 (57.25)

21. Secondary Outcome: Serum Interleukin (IL)-6 Level, Median, From Baseline to Week 48
Description: Serum Interleukin (IL)-6 levels predose at baseline and at subsequent time points after initiation of study drug.
Time Frame: From Baseline to Week 48
Population: as for outcome 9
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 104
pg/mL
  Baseline | 5.21 [0.0 to 15.0] | 4.65 [0.0 to 419.0]
  Week 4: number analyzed (Participants) | 95 | 99
  Week 4 | 5.31 [0.0 to 246.0] | 56.50 [0.0 to 3260.0]
  Week 8: number analyzed (Participants) | 95 | 94
  Week 8 | 5.15 [0.0 to 214.0] | 58.65 [0.0 to 2650.0]
  Week 16: number analyzed (Participants) | 93 | 88
  Week 16 | 5.01 [0.0 to 117.0] | 48.25 [0.0 to 494.0]
  Week 24: number analyzed (Participants) | 85 | 85
  Week 24 | 3.53 [0.0 to 151.0] | 47.90 [0.0 to 286.0]
  Week 36: number analyzed (Participants) | 73 | 83
  Week 36 | 4.01 [0.0 to 107.0] | 46.30 [14.8 to 608.0]
  Week 48: number analyzed (Participants) | 78 | 80
  Week 48 | 3.85 [0.0 to 80.5] | 43.45 [0.0 to 439.0]

22. Secondary Outcome: Serum Interleukin (IL)-6 Level, Mean Change From Baseline to Week 48
Description: Serum Interleukin (IL)-6 levels predose at baseline and at subsequent time points after initiation of study drug.
Time Frame: From Baseline to Week 48
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 104
pg/mL
  Week 4: number analyzed (Participants) | 95 | 99
  Week 4 | 1.11 (28.78) | 130.60 (395.93)
  Week 8: number analyzed (Participants) | 95 | 94
  Week 8 | 2.43 (31.00) | 97.22 (237.43)
  Week 16: number analyzed (Participants) | 93 | 88
  Week 16 | 3.07 (31.71) | 57.10 (62.62)
  Week 24: number analyzed (Participants) | 85 | 85
  Week 24 | 0.13 (30.63) | 53.33 (46.81)
  Week 36: number analyzed (Participants) | 73 | 83
  Week 36 | -3.48 (23.23) | 52.26 (55.81)
  Week 48: number analyzed (Participants) | 78 | 80
  Week 48 | -1.60 (21.54) | 40.01 (29.89)

23. Secondary Outcome: Serum Interleukin (IL)-6 Level, Median Change From Baseline to Week 48
Description: Serum Interleukin (IL)-6 levels predose at baseline and at subsequent time points after initiation of study drug.
Time Frame: From Baseline to Week 48
Population: as for outcome 9
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 104
pg/mL
  Week 4: number analyzed (Participants) | 95 | 99
  Week 4 | -0.12 [-150.0 to 202.7] | 52.41 [-27.4 to 2841.0]
  Week 8: number analyzed (Participants) | 95 | 94
  Week 8 | 0.83 [-148.6 to 210.5] | 52.35 [-9.8 to 2231.0]
  Week 16: number analyzed (Participants) | 93 | 88
  Week 16 | 0.34 [-148.5 to 114.5] | 42.35 [-6.0 to 494.0]
  Week 24: number analyzed (Participants) | 85 | 85
  Week 24 | 0.00 [-148.5 to 144.9] | 41.21 [-8.0 to 284.0]
  Week 36: number analyzed (Participants) | 73 | 83
  Week 36 | 0.00 [-148.2 to 63.3] | 41.20 [0.9 to 474.0]
  Week 48: number analyzed (Participants) | 78 | 80
  Week 48 | 0.00 [-150.0 to 46.0] | 32.96 [-11.8 to 138]

24. Secondary Outcome: Serum Soluble Interleukin (IL)-6 Receptor Level, Mean, From Baseline to Week 48
Description: Serum soluble Interleukin (IL)-6 receptor levels predose at baseline and at subsequent time points after initiation of study drug.
Time Frame: From Baseline to Week 48
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 104
ng/mL
  Baseline: number analyzed (Participants) | 101 | 101
  Baseline | 42.16 (32.41) | 42.22 (14.56)
  Week 4: number analyzed (Participants) | 103 | 102
  Week 4 | 46.07 (73.52) | 486.58 (122.94)
  Week 8: number analyzed (Participants) | 103 | 101
  Week 8 | 45.71 (57.95) | 546.59 (142.58)
  Week 16: number analyzed (Participants) | 102 | 96
  Week 16 | 47.81 (68.22) | 583.87 (164.36)
  Week 24: number analyzed (Participants) | 95 | 95
  Week 24 | 41.35 (15.17) | 587.28 (153.90)
  Week 36: number analyzed (Participants) | 89 | 93
  Week 36 | 38.13 (11.22) | 589.59 (140.63)
  Week 48: number analyzed (Participants) | 91 | 90
  Week 48 | 49.27 (76.97) | 571.48 (167.85)

25. Secondary Outcome: Serum Soluble Interleukin (IL)-6 Receptor Level, Median, From Baseline to Week 48
Description: as for outcome 24
Time Frame: From Baseline to Week 48
Population: as for outcome 9
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 104
ng/mL
  Baseline: number analyzed (Participants) | 101 | 101
  Baseline | 37.10 [17.0 to 340.0] | 39.00 [20.1 to 97.2]
  Week 4: number analyzed (Participants) | 103 | 102
  Week 4 | 38.10 [19.4 to 775.0] | 482.50 [42.0 to 773.0]
  Week 8: number analyzed (Participants) | 103 | 101
  Week 8 | 37.20 [17.6 to 612.0] | 536.00 [30.5 to 873.0]
  Week 16: number analyzed (Participants) | 102 | 96
  Week 16 | 38.95 [20.6 to 711.0] | 589.50 [27.4 to 1290.0]
  Week 24: number analyzed (Participants) | 95 | 95
  Week 24 | 39.30 [19.5 to 99.8] | 590.00 [23.2 to 945.0]
  Week 36: number analyzed (Participants) | 89 | 93
  Week 36 | 36.20 [21.1 to 67.5] | 591.00 [45.4 to 970.0]
  Week 48: number analyzed (Participants) | 91 | 90
  Week 48 | 36.00 [19.2 to 596.0] | 576.50 [23.4 to 973.0]

26. Secondary Outcome: Serum Soluble Interleukin (IL)-6 Receptor Level, Mean Change From Baseline to Week 48
Description: as for outcome 24
Time Frame: From Baseline to Week 48
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 104
ng/mL
  Week 4: number analyzed (Participants) | 99 | 99
  Week 4 | 3.96 (79.00) | 444.23 (120.90)
  Week 8: number analyzed (Participants) | 99 | 98
  Week 8 | 3.31 (65.47) | 501.09 (140.42)
  Week 16: number analyzed (Participants) | 98 | 93
  Week 16 | 6.04 (77.69) | 539.21 (165.63)
  Week 24: number analyzed (Participants) | 91 | 92
  Week 24 | -1.29 (35.46) | 540.98 (152.70)
  Week 36: number analyzed (Participants) | 85 | 90
  Week 36 | -4.31 (35.92) | 544.89 (142.95)
  Week 48: number analyzed (Participants) | 87 | 87
  Week 48 | 7.23 (86.81) | 525.66 (165.53)

27. Secondary Outcome: Serum Soluble Interleukin (IL)-6 Receptor Level, Median Change From Baseline to Week 48
Description: as for outcome 24
Time Frame: From Baseline to Week 48
Population: as for outcome 9
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 104
ng/mL
  Week 4: number analyzed (Participants) | 99 | 99
  Week 4 | 0.20 [-318.4 to 709.5] | 437.80 [-13.4 to 724.3]
  Week 8: number analyzed (Participants) | 99 | 98
  Week 8 | 0.20 [-305.9 to 560.8] | 489.90 [-14.1 to 823.0]
  Week 16: number analyzed (Participants) | 98 | 93
  Week 16 | 0.25 [-316.4 to 679.0] | 542.30 [-28.0 to 1248.7]
  Week 24: number analyzed (Participants) | 91 | 92
  Week 24 | 1.20 [-316.6 to 51.6] | 547.50 [-32.2 to 909.9]
  Week 36: number analyzed (Participants) | 85 | 90
  Week 36 | -0.40 [-315.7 to 24.1] | 541.70 [-26.6 to 942.9]
  Week 48: number analyzed (Participants) | 87 | 87
  Week 48 | -0.70 [-317.9 to 560.2] | 532.20 [-0.4 to 945.9]

28. Secondary Outcome: Serum C-Reactive Protein (CRP) Level, Mean, From Baseline to Week 48
Description: Serum C-Reactive Protein (CRP) levels predose at baseline and at subsequent time points after initiation of study drug.
Time Frame: From Baseline up to Week 48
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 104
mg/L
  Baseline | 7.43 (12.61) | 9.00 (14.76)
  Week 4: number analyzed (Participants) | 102 | 101
  Week 4 | 9.81 (20.79) | 0.85 (2.52)
  Week 24: number analyzed (Participants) | 100 | 97
  Week 24 | 9.89 (13.99) | 0.56 (1.19)
  Week 48: number analyzed (Participants) | 90 | 93
  Week 48 | 7.52 (12.80) | 1.58 (6.22)

29. Secondary Outcome: Serum C-Reactive Protein (CRP) Level, Median, From Baseline to Week 48
Description: Serum C-Reactive Protein (CRP) levels predose at baseline and at subsequent time points after initiation of study drug.
Time Frame: From Baseline up to Week 48
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 104
mg/L
  Baseline | 3.82 [1.19 to 8.69] | 4.05 [1.30 to 9.48]
  Week 4: number analyzed (Participants) | 102 | 101
  Week 4 | 3.71 [1.27 to 8.83] | 0.20 [0.20 to 0.50]
  Week 24: number analyzed (Participants) | 100 | 97
  Week 24 | 4.15 [1.43 to 13.10] | 0.20 [0.20 to 0.47]
  Week 48: number analyzed (Participants) | 90 | 93
  Week 48 | 3.67 [1.26 to 7.78] | 0.20 [0.20 to 0.59]

30. Secondary Outcome: Serum Tocilizumab Concentration, Mean, From Baseline to Week 48
Description: Predose observed serum TCZ concentration at baseline and at specified timepoints thereafter
Time Frame: From Baseline to Week 48
Population: The PK population includes all patients who received at least one TCZ injection and had at least one PK sample with detectable results.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Double-Blind Tocilizumab
Number analyzed (Participants) | 103
ug/mL
  Baseline: number analyzed (Participants) | 100
  Baseline | 0.00 (0.03)
  Week 4: number analyzed (Participants) | 102
  Week 4 | 30.92 (15.24)
  Week 8: number analyzed (Participants) | 100
  Week 8 | 41.82 (17.66)
  Week 16: number analyzed (Participants) | 93
  Week 16 | 50.98 (23.33)
  Week 24: number analyzed (Participants) | 93
  Week 24 | 54.34 (26.24)
  Week 36: number analyzed (Participants) | 91
  Week 36 | 53.55 (29.25)
  Week 48: number analyzed (Participants) | 88
  Week 48 | 54.67 (29.79)

31. Secondary Outcome: Serum Tocilizumab Concentration, Median, From Baseline to Week 48
Description: Predose observed serum TCZ concentration at baseline and at specified timepoints thereafter
Time Frame: From Baseline to Week 48
Population: as for outcome 30
Measure: Median (Full Range); unit: ug/mL
Arm/Group | Double-Blind Tocilizumab
Number analyzed (Participants) | 103
ug/mL
  Baseline: number analyzed (Participants) | 100
  Baseline | 0.00 [0.0 to 0.2]
  Week 4: number analyzed (Participants) | 102
  Week 4 | 28.70 [0.4 to 86.8]
  Week 8: number analyzed (Participants) | 100
  Week 8 | 39.25 [8.3 to 97.6]
  Week 16: number analyzed (Participants) | 93
  Week 16 | 47.40 [9.5 to 120.0]
  Week 24: number analyzed (Participants) | 93
  Week 24 | 52.60 [7.6 to 117.0]
  Week 36: number analyzed (Participants) | 91
  Week 36 | 52.50 [4.0 to 138.0]
  Week 48: number analyzed (Participants) | 88
  Week 48 | 52.10 [0.4 to 145.0]

32. Secondary Outcome: Correlation Between Low Serum Tocilizumab Exposure and Mean Modified Rodnan Skin Score (mRSS) From Baseline to Week 48
Description: In order to characterize exposure-efficacy relationships, mRSS scores are summarized based on TCZ exposure tertiles (high, medium, and low exposures) in the active treatment group and compared to placebo patients. Low Exposure = 0-<41 ug/ml, Medium = 41-<=61.1 ug/ml, High = 61.1-<=145 ug/ml.
Time Frame: From Baseline to Week 48
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 30
Units on a scale
  Baseline | 20.4 (6.95) | 20.3 (5.56)
  Week 8: number analyzed (Participants) | 102 | 30
  Week 8 | 18.6 (7.78) | 17.9 (5.84)
  Week 16: number analyzed (Participants) | 101 | 29
  Week 16 | 17.9 (8.71) | 16.2 (5.58)
  Week 24: number analyzed (Participants) | 99 | 30
  Week 24 | 16.9 (9.38) | 14.7 (5.61)
  Week 36: number analyzed (Participants) | 94 | 30
  Week 36 | 16.2 (10.24) | 13.2 (4.97)
  Week 48: number analyzed (Participants) | 92 | 30
  Week 48 | 14.8 (9.89) | 12.2 (6.03)

33. Secondary Outcome: Correlation Between Low Serum Tocilizumab Exposure and Median Modified Rodnan Skin Score (mRSS) From Baseline to Week 48
Description: as for outcome 32
Time Frame: From Baseline to Week 48
Population: as for outcome 9
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 30
Units on a scale
  Baseline | 19.0 [10 to 40] | 20.0 [11 to 31]
  Week 8: number analyzed (Participants) | 102 | 30
  Week 8 | 18.0 [4 to 43] | 16.0 [9 to 34]
  Week 16: number analyzed (Participants) | 101 | 29
  Week 16 | 17.0 [0 to 38] | 15.0 [8 to 30]
  Week 24: number analyzed (Participants) | 99 | 30
  Week 24 | 16.0 [0 to 42] | 14.0 [6 to 29]
  Week 36: number analyzed (Participants) | 94 | 30
  Week 36 | 14.0 [0 to 47] | 13.5 [5 to 27]
  Week 48: number analyzed (Participants) | 92 | 30
  Week 48 | 14.0 [0 to 43] | 12.5 [2 to 30]

34. Secondary Outcome: Correlation Between Medium Serum Tocilizumab Exposure and Mean Modified Rodnan Skin Score (mRSS) From Baseline to Week 48
Description: as for outcome 32
Time Frame: From Baseline to Week 48
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 29
Units on a scale
  Baseline | 20.4 (6.95) | 19.1 (6.24)
  Week 8: number analyzed (Participants) | 102 | 29
  Week 8 | 18.6 (7.78) | 17.2 (6.17)
  Week 16: number analyzed (Participants) | 101 | 29
  Week 16 | 17.9 (8.71) | 16.2 (6.10)
  Week 24: number analyzed (Participants) | 99 | 29
  Week 24 | 16.9 (9.38) | 14.6 (6.66)
  Week 36: number analyzed (Participants) | 94 | 28
  Week 36 | 16.2 (10.24) | 13.4 (6.20)
  Week 48: number analyzed (Participants) | 92 | 29
  Week 48 | 14.8 (9.89) | 11.6 (5.72)

35. Secondary Outcome: Correlation Between Medium Serum Tocilizumab Exposure and Median Modified Rodnan Skin Score (mRSS) From Baseline to Week 48
Description: as for outcome 32
Time Frame: From Baseline to Week 48
Population: as for outcome 9
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 29
Units on a scale
  Baseline | 19.0 [10 to 40] | 18.0 [10 to 35]
  Week 8: number analyzed (Participants) | 102 | 29
  Week 8 | 18.0 [4 to 43] | 17.0 [5 to 31]
  Week 16: number analyzed (Participants) | 101 | 29
  Week 16 | 17.0 [0 to 38] | 16.0 [5 to 27]
  Week 24: number analyzed (Participants) | 99 | 29
  Week 24 | 16.0 [0 to 42] | 14.0 [3 to 28]
  Week 36: number analyzed (Participants) | 94 | 28
  Week 36 | 14.0 [0 to 47] | 13.0 [2 to 25]
  Week 48: number analyzed (Participants) | 92 | 29
  Week 48 | 14.0 [0 to 43] | 11.0 [0 to 24]

36. Secondary Outcome: Correlation Between High Serum Tocilizumab Exposure and Mean Modified Rodnan Skin Score (mRSS) From Baseline to Week 48
Description: as for outcome 32
Time Frame: From Baseline to Week 48
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 29
Units on a scale
  Baseline | 20.4 (6.95) | 19.8 (6.82)
  Week 8: number analyzed (Participants) | 102 | 28
  Week 8 | 18.6 (7.78) | 17.9 (7.35)
  Week 16: number analyzed (Participants) | 101 | 29
  Week 16 | 17.9 (8.71) | 16.7 (7.31)
  Week 24: number analyzed (Participants) | 99 | 29
  Week 24 | 16.9 (9.38) | 15.6 (7.50)
  Week 36: number analyzed (Participants) | 94 | 28
  Week 36 | 16.2 (10.24) | 13.7 (7.07)
  Week 48: number analyzed (Participants) | 92 | 29
  Week 48 | 14.8 (9.89) | 12.8 (7.20)

37. Secondary Outcome: Correlation Between High Serum Tocilizumab Exposure and Median Modified Rodnan Skin Score (mRSS) From Baseline to Week 48
Description: as for outcome 32
Time Frame: From Baseline to Week 48
Population: as for outcome 9
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 106 | 29
Units on a scale
  Baseline | 19.0 [10 to 40] | 19.0 [11 to 33]
  Week 8: number analyzed (Participants) | 102 | 28
  Week 8 | 18.0 [4 to 43] | 17.5 [5 to 32]
  Week 16: number analyzed (Participants) | 101 | 29
  Week 16 | 17.0 [0 to 38] | 15.0 [6 to 33]
  Week 24: number analyzed (Participants) | 99 | 29
  Week 24 | 16.0 [0 to 42] | 15.0 [2 to 31]
  Week 36: number analyzed (Participants) | 94 | 28
  Week 36 | 14.0 [0 to 47] | 11.0 [4 to 30]
  Week 48: number analyzed (Participants) | 92 | 29
  Week 48 | 14.0 [0 to 43] | 11.0 [4 to 34]

38. Secondary Outcome: Change in Mean Modified Rodnan Skin Score (mRSS) at Low, Medium and High Serum Tocilizumab Exposure From Baseline to Week 48
Description: as for outcome 32
Time Frame: From Baseline to Week 48
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 92 | 30
Units on a scale
  Low Exposure | -5.3 (7.77) | -8.0 (5.85)
  Medium Exposure: number analyzed (Participants) | 92 | 29
  Medium Exposure | -5.3 (7.77) | -7.5 (5.06)
  High Exposure: number analyzed (Participants) | 92 | 29
  High Exposure | -5.3 (7.77) | -7.0 (6.26)

39. Secondary Outcome: Change in Median Modified Rodnan Skin Score (mRSS), at Low, Medium and High Serum Tocilizumab Exposure From Baseline to Week 48
Description: as for outcome 32
Time Frame: From Baseline to Week 48
Population: as for outcome 9
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 92 | 30
Units on a scale
  Low Exposure | -5.5 [-25 to 22] | -8.0 [-19 to 4]
  Medium Exposure | -5.5 [-25 to 22] | -7.0 [-18 to 2]
  High Exposure | -5.5 [-25 to 22] | -6.0 [-20 to 6]

40. Secondary Outcome: Change in Mean Percent Predicted Forced Vital Capacity (ppFVC), at Low, Medium and High Serum Tocilizumab Exposure From Baseline to Week 48
Description: In order to characterize exposure-efficacy relationships, ppFVC scores are summarized based on TCZ exposure tertiles (high, medium, and low exposures) in the active treatment group and compared to placebo patients. Low Exposure = 0-<41 ug/ml, Medium = 41-<=61.1 ug/ml, High = 61.1-<=145 ug/ml.
Time Frame: From Baseline to Week 48
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 91 | 29
Percent
  Low Exposure: number analyzed (Participants) | 91 | 28
  Low Exposure | -4.264 (8.155) | 0.144 (6.474)
  Medium Exposure: number analyzed (Participants) | 91 | 28
  Medium Exposure | -4.264 (8.155) | -0.161 (6.440)
  High Exposure | -4.264 (8.155) | -0.297 (7.895)

41. Secondary Outcome: Change in Median Percent Predicted Forced Vital Capacity (ppFVC), at Low, Medium and High Serum Tocilizumab Exposure From Baseline to Week 48
Description: as for outcome 40
Time Frame: From Baseline to Week 48
Population: as for outcome 9
Measure: Median (Full Range); unit: Percent
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab
Number analyzed (Participants) | 91 | 29
Percent
  Low Exposure: number analyzed (Participants) | 91 | 28
  Low Exposure | -3.910 [-31.47 to 13.47] | 0.525 [-14.25 to 11.38]
  Medium Exposure: number analyzed (Participants) | 91 | 28
  Medium Exposure | -3.910 [-31.47 to 13.47] | -1.600 [-13.83 to 17.00]
  High Exposure | -3.910 [-31.47 to 13.47] | 0.000 [-10.55 to 19.69]

42. Secondary Outcome: Summary of Adverse Events Up to Week 96
Description: Summary of key safety results including Adverse Events of Special Interest (AESI). All adverse events categorized according to MedDRA version 21.1. NMSC = Non-Melanoma Skin Cancer
Time Frame: Up to Week 96
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Groups:
- Placebo, Then Tocilizumab Open Label: Participants who received placebo during the double blind period from Baseline to Week 48, received tocilizumab from Week 48 to Week 96.
- Tocilizumab, Then Tocilizumab Open Label: Participants who received tocilizumab during the double blind period from Baseline to Week 48, received tocilizumab from Week 48 to Week 96.
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab | Placebo, Then Tocilizumab Open Label | Tocilizumab, Then Tocilizumab Open Label
Number analyzed (Participants) | 106 | 104 | 89 | 92
Percentage of participants
  At least one Adverse Event (AE) | 77.4 | 85.6 | 77.5 | 71.7
  Withdrawn from study due to an AE | 12.3 | 6.7 | 1.1 | 1.1
  Fatal AE | 2.8 | 1.0 | 1.1 | 1.1
  Serious Adverse Events (SAEs) | 17.0 | 12.5 | 7.9 | 10.9
  SAE leading to withdrawal from treatment | 5.7 | 4.8 | 1.1 | 1.1
  SAE leading to dose modification/interruption | 5.7 | 2.9 | 4.5 | 3.3
  SAE related to study drug | 6.6 | 1.0 | 3.4 | 3.3
  AE leading to withdrawal from treatment | 12.3 | 6.7 | 1.1 | 1.1
  AE leading to dose modification/interruption | 26.4 | 19.2 | 28.1 | 22.8
  AE related to study drug | 34.0 | 46.2 | 33.7 | 34.8
  Related AE leading to withdrawal from treatment | 1.9 | 1.0 | 1.1 | 1.1
  Related AE with dose modification/interruption | 17.0 | 11.5 | 12.4 | 14.1
  Serious Infections and Infestations AEs | 6.6 | 1.9 | 3.4 | 1.1
  Infections and Infestations AEs | 50.0 | 52.9 | 46.1 | 39.1
  Opportunistic Infections AEs | 0.9 | 1.0 | 0 | 1.1
  Malignancy AEs | 0.9 | 1.9 | 0 | 1.1
  Malignancy AEs (excluding NMSC) | 0.9 | 1.9 | 0 | 1.1
  Serious Hepatic AEs | 0 | 0 | 0 | 0
  Serious Stroke AEs | 0 | 0 | 0 | 0
  Serious Myocardial Infarction AEs | 1.9 | 0 | 0 | 0
  Anaphylactic Reaction AEs | 0 | 0 | 0 | 0
  Anaphylactic Reaction AEs (Sampson's Criteria) | 0 | 0 | 0 | 0
  Serious Gastrointestinal Perforation AEs | 0 | 0 | 0 | 0
  Serious Bleeding AEs | 0.9 | 0 | 0 | 0
  Serious Demyelinating AEs | 0 | 0 | 0 | 0

43. Secondary Outcome: Incidence and Severity of Adverse Events Up to Week 96
Description: Adverse events according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) severity grade: 1 = mild, 2 = moderate, 3 = severe and/or requiring medical intervention but not life-threatening, 4 = life-threatening consequences, and 5 = death.
Time Frame: Up to Week 96
Population: as for outcome 9
Measure: Number; unit: Number of participants
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab | Placebo, Then Tocilizumab Open Label | Tocilizumab, Then Tocilizumab Open Label
Number analyzed (Participants) | 106 | 104 | 89 | 92
Number of participants
  Grade 1 | 61 | 78 | 60 | 53
  Grade 2 | 63 | 53 | 41 | 35
  Grade 3 | 21 | 18 | 9 | 8
  Grade 4 | 7 | 0 | 4 | 5
  Grade 5 | 3 | 1 | 1 | 1

44. Secondary Outcome: Number of Participants With Adverse Events Leading to Death Up to Week 96
Time Frame: Up to Week 96
Population: as for outcome 9
Measure: Number; unit: Number of participants
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab | Placebo, Then Tocilizumab Open Label | Tocilizumab, Then Tocilizumab Open Label
Number analyzed (Participants) | 106 | 104 | 89 | 92
Number of participants
  CARDIAC FAILURE CHRONIC | 1 | 0 | 0 | 0
  MYOCARDITIS | 1 | 0 | 0 | 0
  MYOCARDIAL INFARCTION | 1 | 0 | 0 | 0
  DEATH | 0 | 1 | 0 | 0
  BRAIN INJURY | 0 | 0 | 1 | 0
  PULMONARY HYPERTENSION | 0 | 0 | 0 | 1

45. Secondary Outcome: Percentage of Participants With Change in Digital Ulcer Count at Week 96
Description: as for outcome 14
Time Frame: From Baseline to Week 96
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab | Placebo, Then Tocilizumab Open Label | Tocilizumab, Then Tocilizumab Open Label
Number analyzed (Participants) | 106 | 104 | 89 | 92
Percentage of participants
  No change | 0 | 0 | 91.1 | 83.3
  Increase by 1 | 0 | 0 | 0 | 4.8
  Increase by 2 | 0 | 0 | 0 | 1.2
  Increase by 3 | 0 | 0 | 0 | 1.2
  Increase by 4 | 0 | 0 | 0 | 0
  Increase by >4 | 0 | 0 | 0 | 1.2
  Decrease by 1 | 0 | 0 | 3.8 | 4.8
  Decrease by 2 | 0 | 0 | 2.5 | 0
  Decrease by 3 | 0 | 0 | 1.3 | 1.2
  Decrease by 4 | 0 | 0 | 1.3 | 1.2
  Decrease by >4 | 0 | 0 | 0 | 0
  Baseline missing | 0 | 0 | 0 | 1.2

46. Secondary Outcome: Percentage of Participants With Positive Anti-Tocilizumab Assay Post-Baseline From Week 48 to 96
Description: Reported were the percentage of participants with post-baseline treatment-induced anti-TCZ antibodies. Positive samples underwent additional analyses: a neutralizing assay for the ability to inhibit the activity of TCZ and a test for anti -TCZ of the IgE isotype.
Time Frame: Open-label period from Week 48 to 96
Population: Safety population: received at least one dose of study drug and provide data from at least one post dose safety assessment. Only samples from the Double Blind TCZ, then Open Label TCZ were measured by the lab after week 48. Data for the Double Blind Period were reported at the time of Primary Results disclosure up to Week 48.
Measure: Number; unit: Percentage of Participants
Groups:
- Tocilizumab, Then Tocilizumab Open Label: Participants who received tocilizumab during the double blind period from Baseline to Week 47, received tocilizumab from Week 48 to Week 96.
Arm/Group | Tocilizumab, Then Tocilizumab Open Label
Number analyzed (Participants) | 92
Percentage of Participants
  Treatment-Induced Anti-TCZ Antibodies | 0.0
  Anti-TCZ Antibodies of Neutralizing Potential | 0.0
  Anti-TCZ Antibodies of IgE | 0.0

47. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR) Up to Week 96
Description: as for outcome 18
Time Frame: Up to Week 96
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab | Placebo, Then Tocilizumab Open Label | Tocilizumab, Then Tocilizumab Open Label
Number analyzed (Participants) | 103 | 100 | 82 | 89
mm/hr
  Baseline: number analyzed (Participants) | 103 | 100 | 0 | 0
  Baseline | 34.72 (18.49) | 34.83 (16.29) |  |
  Week 4: number analyzed (Participants) | 96 | 98 | 0 | 0
  Week 4 | 31.38 (19.00) | 14.29 (12.98) |  |
  Week 24: number analyzed (Participants) | 98 | 94 | 0 | 0
  Week 24 | 28.49 (20.86) | 8.46 (8.63) |  |
  Week 48: number analyzed (Participants) | 91 | 93 | 0 | 0
  Week 48 | 26.23 (18.53) | 10.89 (15.39) |  |
  Week 72: number analyzed (Participants) | 0 | 0 | 82 | 89
  Week 72 |  |  | 9.54 (9.47) | 8.29 (10.13)
  Week 96: number analyzed (Participants) | 0 | 0 | 79 | 85
  Week 96 |  |  | 9.67 (8.67) | 8.06 (8.86)

48. Secondary Outcome: Serum Interleukin (IL)-6 Level, Mean, From Baseline to Week 96
Description: Serum Interleukin (IL)-6 levels predose at baseline and at subsequent time points after initiation of study drug.
Time Frame: Up to Week 96
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab | Placebo, Then Tocilizumab Open Label | Tocilizumab, Then Tocilizumab Open Label
Number analyzed (Participants) | 106 | 104 | 79 | 79
pg/mL
  Baseline: number analyzed (Participants) | 106 | 104 | 0 | 0
  Baseline | 11.85 (19.73) | 13.86 (43.78) |  |
  Week 4: number analyzed (Participants) | 95 | 98 | 0 | 0
  Week 4 | 13.41 (29.98) | 144.75 (429.14) |  |
  Week 8: number analyzed (Participants) | 95 | 94 | 0 | 0
  Week 8 | 14.21 (26.82) | 111.44 (280.34) |  |
  Week 16: number analyzed (Participants) | 93 | 88 | 0 | 0
  Week 16 | 15.40 (24.26) | 66.20 (70.50) |  |
  Week 24: number analyzed (Participants) | 85 | 85 | 0 | 0
  Week 24 | 11.81 (24.05) | 62.74 (53.40) |  |
  Week 36: number analyzed (Participants) | 73 | 83 | 0 | 0
  Week 36 | 9.32 (15.23) | 62.15 (68.08) |  |
  Week 48: number analyzed (Participants) | 81 | 82 | 0 | 0
  Week 48 | 9.10 (14.88) | 53.34 (56.80) |  |
  Week 96: number analyzed (Participants) | 0 | 0 | 79 | 79
  Week 96 |  |  | 62.60 (57.21) | 52.03 (46.51)

49. Secondary Outcome: Serum Soluble Interleukin (IL)-6 Receptor Level, Mean, Up to Week 96
Description: as for outcome 24
Time Frame: Up to Week 96
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab | Placebo, Then Tocilizumab Open Label | Tocilizumab, Then Tocilizumab Open Label
Number analyzed (Participants) | 103 | 102 | 79 | 85
ng/mL
  Baseline: number analyzed (Participants) | 100 | 102 | 0 | 0
  Baseline | 42.23 (32.56) | 42.15 (14.50) |  |
  Week 4: number analyzed (Participants) | 103 | 101 | 0 | 0
  Week 4 | 46.07 (73.52) | 487.70 (123.02) |  |
  Week 8: number analyzed (Participants) | 103 | 101 | 0 | 0
  Week 8 | 45.71 (57.95) | 546.59 (142.58) |  |
  Week 16: number analyzed (Participants) | 102 | 96 | 0 | 0
  Week 16 | 47.81 (68.22) | 583.87 (164.36) |  |
  Week 24: number analyzed (Participants) | 95 | 95 | 0 | 0
  Week 24 | 41.35 (15.17) | 587.28 (153.90) |  |
  Week 36: number analyzed (Participants) | 89 | 93 | 0 | 0
  Week 36 | 38.13 (11.22) | 589.59 (140.63) |  |
  Week 48: number analyzed (Participants) | 93 | 92 | 0 | 0
  Week 48 | 49.51 (76.17) | 566.49 (175.25) |  |
  Week 96: number analyzed (Participants) | 0 | 0 | 79 | 85
  Week 96 |  |  | 558.38 (256.86) | 565.31 (159.82)

50. Secondary Outcome: Serum C-Reactive Protein (CRP) Level, Mean, Up to Week 96
Description: Serum C-Reactive Protein (CRP) levels predose at baseline and at subsequent time points after initiation of study drug.
Time Frame: From Baseline up to Week 96
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab | Placebo, Then Tocilizumab Open Label | Tocilizumab, Then Tocilizumab Open Label
Number analyzed (Participants) | 106 | 104 | 83 | 90
mg/L
  Baseline: number analyzed (Participants) | 106 | 104 | 0 | 0
  Baseline | 7.42 (12.62) | 8.99 (14.76) |  |
  Week 4: number analyzed (Participants) | 103 | 103 | 0 | 0
  Week 4 | 10.05 (20.82) | 0.85 (2.50) |  |
  Week 24: number analyzed (Participants) | 100 | 97 | 0 | 0
  Week 24 | 9.89 (13.99) | 0.56 (1.19) |  |
  Week 48: number analyzed (Participants) | 93 | 96 | 0 | 0
  Week 48 | 7.40 (12.62) | 1.75 (6.43) |  |
  Week 72: number analyzed (Participants) | 0 | 0 | 82 | 90
  Week 72 |  |  | 0.57 (0.80) | 0.92 (3.61)
  Week 96: number analyzed (Participants) | 0 | 0 | 83 | 86
  Week 96 |  |  | 0.90 (2.73) | 0.97 (5.08)

51. Secondary Outcome: Serum Tocilizumab Concentration, Mean, Up to Week 96
Description: Predose observed serum TCZ concentration at baseline and at specified timepoints thereafter
Time Frame: Up to Week 96
Population: The PK population included all participants who received at least one TCZ injection and had at least one PK sample with detectable results. Only samples from the Double Blind TCZ, then Open Label TCZ were measured by the lab after week 48. Data for the Double Blind Period were reported at the time of Primary Results disclosure up to Week 48.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Double-Blind Tocilizumab, Then Open Label Tocilizumab
Number analyzed (Participants) | 101
ug/mL
  Baseline | 0.00 (0.03)
  Week 4 | 30.76 (15.23)
  Week 8: number analyzed (Participants) | 100
  Week 8 | 41.82 (17.66)
  Week 16: number analyzed (Participants) | 93
  Week 16 | 50.98 (23.33)
  Week 24: number analyzed (Participants) | 93
  Week 24 | 54.34 (26.24)
  Week 36: number analyzed (Participants) | 91
  Week 36 | 53.55 (29.25)
  Week 48: number analyzed (Participants) | 89
  Week 48 | 54.87 (29.69)
  Week 96: number analyzed (Participants) | 82
  Week 96 | 49.99 (26.19)

ADVERSE EVENTS:
Time Frame: Up to Week 96
Description: The analysis was conducted in the safety population i.e. received at least one dose of study drug and provide data from at least one post dose safety assessment.
Arm/Group | Double-Blind Placebo | Double-Blind Tocilizumab | Placebo, Then Tocilizumab Open Label | Tocilizumab, Then Tocilizumab Open Label
All-Cause Mortality (participants affected / at risk) | 3/106 | 1/104 | 1/89 | 1/92
Serious Adverse Events (participants affected / at risk) | 18/106 | 13/104 | 7/89 | 10/92
Other Adverse Events (participants affected / at risk) | 59/106 | 60/104 | 46/89 | 28/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-Blind Placebo (N=106) | Double-Blind Tocilizumab (N=104) | Placebo, Then Tocilizumab Open Label (N=89) | Tocilizumab, Then Tocilizumab Open Label (N=92)
ANAEMIA MEGALOBLASTIC (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LYMPHADENOPATHY MEDIASTINAL (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ARRHYTHMIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CARDIAC TAMPONADE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONGESTIVE CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MICROVASCULAR CORONARY ARTERY DISEASE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MYOCARDITIS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RETINAL VEIN THROMBOSIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTRITIS EROSIVE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ILEUS PARALYTIC (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RECTAL PROLAPSE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DEATH (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INFECTED SKIN ULCER (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INFECTIVE TENOSYNOVITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OSTEOMYELITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTITIS MEDIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PELVIC INFLAMMATORY DISEASE (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
PYELONEPHRITIS CHRONIC (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
SOFT TISSUE INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
WOUND INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LIMB TRAUMATIC AMPUTATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SPINAL CORD INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
WEIGHT DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
JOINT STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SCLERODERMA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TENOSYNOVITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TRIGGER FINGER (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BENIGN BONE NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
BRAIN INJURY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ADJUSTMENT DISORDER (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SCLERODERMA RENAL CRISIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DIGITAL PITTING SCAR (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-Blind Placebo (N=106) | Double-Blind Tocilizumab (N=104) | Placebo, Then Tocilizumab Open Label (N=89) | Tocilizumab, Then Tocilizumab Open Label (N=92)
ANAEMIA (Blood and lymphatic system disorders) | 6 (6) | 2 (2) | 1 (1) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 7 (7) | 6 (7) | 6 (7) | 5 (5)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 6 (6) | 4 (4) | 8 (8) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 6 (6) | 3 (3) | 2 (2) | 1 (1)
FATIGUE (General disorders) | 7 (8) | 8 (9) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 2 (2) | 7 (7) | 0 (0) | 3 (3)
NASOPHARYNGITIS (Infections and infestations) | 8 (9) | 13 (14) | 9 (10) | 4 (4)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 11 (15) | 12 (13) | 10 (16) | 4 (5)
URINARY TRACT INFECTION (Infections and infestations) | 10 (14) | 5 (5) | 7 (8) | 1 (1)
WEIGHT DECREASED (Investigations) | 6 (6) | 2 (2) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 14 (15) | 12 (14) | 3 (3) | 5 (5)
HEADACHE (Nervous system disorders) | 6 (6) | 3 (3) | 1 (1) | 1 (2)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 2 (2) | 1 (1) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 4 (5) | 6 (6) | 2 (3) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 7 (8) | 2 (2) | 3 (3) | 2 (2)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 12 (22) | 15 (28) | 16 (28) | 11 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-01-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT02453256/SAP_001.pdf
  • Study Protocol (2017-05-05): https://cdn.clinicaltrials.gov/large-docs/56/NCT02453256/Prot_002.pdf